# The GlaxoSmithKline group of companies

205801

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for a Phase II, Randomized,
Open-label Platform Trial Utilizing a Master Protocol to Study
Novel Regimens Versus Standard of Care Treatment in
NSCLC Participants

Compound Number : GSK3359609

Effective Date : Refer to Document Date

#### **Description:**

- The purpose of this RAP is to describe the planned final analyses and outputs for each substudy in the Clinical Study Report (CSR) for 205801. Separate CSRs will be produced for each substudy.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

# RAP Author(s):



Copyright 2021 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited

# The GlaxoSmithKline group of companies

205801

# **RAP Team Review Confirmations (Method: E-mail)**

| Reviewer | Date |
|---------------------------------------------------------|-------------|
| PPD Clinical Investigation Lead (Oncology, Clinical) | 03-Mar-2021 |
| PPD Safety Lead (SMG, Pharma Safety) | 02-Mar-2021 |
| PPD Physician, ICOS (Oncology) | 05-Mar-2021 |
| PPD Study Data Manager (SDM), Clinical Data Management | 03-Mar-2021 |
| PPD Patients Centered Outcomes, VEO | 04-Mar-2021 |
| PPD Programming Leader (Oncology, Clinical Programming) | 02-Mar-2021 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | |
|----------|----------------------------------|
| PPD | |
| PPD | (Biostatistics, GSK) |
| PPD | |
| PPD | Programming (Biostatistics, GSK) |

# **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| TA | ABLE OF CONTENTS | 3 |
| 1. | INTRODUCTION | 7 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 7 |
| ۷. | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. Study Objective(s) and Endpoint(s) | |
| | 2.3. Study Design | |
| | 2.4. Statistical Hypotheses / Statistical Analyses | 12 |
| | 2.4.1. Hypothesis | |
| | 2.4.2. Sample Size | |
| 3. | PLANNED ANALYSES | 15 |
| | 3.1. Interim Analyses | 15 |
| | 3.1.1. Interim Analyses for Overall Survival (OS) | 15 |
| | 3.2. Primary and Final Analyses | 16 |
| 4. | ANALYSIS POPULATIONS | 17 |
| | 4.1. Protocol Deviations | |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDL | ING |
| | | 18 |
| | 5.1. Study Treatment & Sub-group Display Descriptors | |
| | 5.2. Baseline Definitions | |
| | 5.3. Multicentre Studies | |
| | 5.4. Examination of Covariates, Other Strata and Subgroups | |
| | 5.4.1. Covariates and Other Strata | |
| | 5.4.2. Examination of Subgroups | |
| | 5.5. Multiple Comparisons and Multiplicity | |
| | 5.6. Other Considerations for Data Analyses and Data Handlir Conventions | |
| 6. | STUDY POPULATION ANALYSES | 21 |
| 0. | 6.1. Overview of Planned Study Population Analyses | |
| | 6.2. Disposition of Subjects | |
| | 6.3. Demographic and Baseline Characteristics | ۱ کــــــــــــــــــــــــــــــــــــ |
| | 6.4. Prior Medical Condition and Disease Characteristics | |
| | 6.5. Prior and Subsequent Anti-cancer Therapy | |
| | 6.6. Concomitant Medications | |
| 7. | EFFICACY ANALYSES | 24 |
| | 7.1. Primary Efficacy Analyses | |
| | 7.1.1. Endpoint / Variables | |
| | 7.1.2. Summary Measure | |
| | 7.1.3. Population of Interest | |
| | 7.1.4. Strategy for Intercurrent (Post-Randomization) E | events24 |
| | 7.1.5. Statistical Analyses / Methods | |
| | 7.2 Secondary Efficacy Analyses | 30 |

205801

| | | 7.2.1. | Endpoint / Variables | 30 |
|---|---|---|---|---|
| | | 7.2.2. | Summary Measure | |
| | | 7.2.3. | Population of Interest | |
| | | 7.2.4. | Statistical Analyses / Methods | |
| | | | 7.2.4.1. Statistical Methodology Specification | |
| 8. | SAFE | Τν ΔΝΔΙ Ν | YSES | 38 |
| 0. | 8.1. | | f Exposure | |
| | 8.2. | | Events Analyses | |
| | 8.3. | | Events of Special Interest Analyses | |
| | 8.4. | | and Serious Adverse Events | |
| | 8.5. | | Events Leading to Discontinuation of Study Treatment | |
| | | and/or W | /ithdrawal from the Study and Other Significant Adverse | |
| | | | ······································ | 47 |
| | 8.6. | | cies | |
| | 8.7. | | _aboratory Analyses | |
| | 8.8. | Liver Fur | nction Analyses | 49 |
| | 8.9. | | afety Analyses | |
| 9. | | | NETIC ANALYSES | |
| | 9.1. | | Pharmacokinetic Analyses | |
| | 9.2. | | ry Pharmacokinetic Analyses | 52 |
| | | 9.2.1. | Endpoint / Variables | |
| | | | 9.2.1.1. Drug Concentration Measures | |
| | | | 9.2.1.2. Derived Pharmacokinetic Parameters | |
| | | 9.2.2. | Summary Measure | |
| | | 9.2.3. | Population of Interest | |
| | | 9.2.4. | Strategy for Intercurrent (Post-Randomization) Events | 53 |
| 10 | SECO | NDARY A | NALYSES | 53 |
| | 10.1. | | genicity Analyses | |
| | 10.2. | | Reported Outcomes | |
| | | 10.2.1. | Endpoint / Variables | |
| | | 10.2.2. | Population of Interest | |
| | | 10.2.3. | Statistical Measures | E 4 |
| | | | 10.2.3.1. Summary Measure | 54 |
| 11. | REFE | RENCES. | | 57 |
| 12 | APPE | NDICES | | 59 |
| 12. | 12.1. | | x 1: Protocol Deviation Management and Definitions for Per | 00 |
| | | | Population | 59 |
| | 12.2. | Appendix | x 2: Schedule of Activities | 60 |
| | 12.2. | 12.2.1. | | 60 |
| | 12.3. | | x 3: Assessment Windows | |
| | 12.4. | | x 4: Study Phases and Treatment Emergent Adverse | |
| | | | | 62 |
| | | 12.4.1. | | |
| | | | 12.4.1.1. Study Phases for Concomitant Medication | |
| | | 12.4.2. | Treatment Emergent Flag for Adverse Events | |
| | 12.5. | | x 5: Data Display Standards & Handling Conventions | 64 |
| | | 1251 | Reporting Process | 64 |

| | | | | 205801 |
|---|---|---|---|---|
| | | 12.5.2. | Reporting Standards | 64 |
| | | 12.5.3. | Reporting Standards for Pharmacokinetic | |
| | 12.6. | | x 6: Derived and Transformed Data | |
| | | 12.6.1. | General | |
| | | 12.6.2. | Study Population | |
| | | 12.6.3. | Safety | |
| | | 12.6.4. | | 68 |
| | | | CCI | |
| | 40.7 | A | . 7. Dan antion Otan dands for Mission Data | 70 |
| | 12.7. | | x 7: Reporting Standards for Missing Data | /6 |
| | | 12.7.1. | Tomatara Transaction | |
| | | 12.7.2. | Handling of Missing Data | |
| | 12.8. | Annondi | 12.7.2.1. Handling of Missing and Partial Dates | |
| | 12.0. | | x 8: Values of Potential Clinical Importancex 9: Abbreviations & Trade Marks | |
| | 12.9. | | Abbreviations | |
| | | 12.9.1. | Trademarks | |
| | 12 10 | | x 10: List of Data Displays | |
| | 12.10. | | Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverables | |
| | | | Study Population Tables | |
| | | | Efficacy Tables | |
| | | | Efficacy Figures | |
| | | | Safety Tables | |
| | | | Safety Figures | |
| | | 12.10.9. | Pharmacokinetic Tables | 99 |
| | | | .Pharmacokinetic Figures | |
| | | 12.10.11 | .Patient Reported Outcomes Tables | 101 |
| | | | .Patient Reported Outcomes Figures | |
| | | 12.10.13 | .ICH Listings | 105 |
| | | 12.10.14 | .Non-ICH Listings | 110 |
| | 12.11. | Appendix | x 11: Example Mock Shells for Data Displays | 111 |
| | 12.12. | Appendix | x 12: SDAC REPORTING PLAN | 112 |
| 13. | | | N | |
| | 13.1. | | ces to External Documents | |
| | 13.2. | | EW OF ANALYSES SPECIFIED IN THE IDMC CHARTER | |
| | 13.3. | | AL SDAC REPORTING CONVENTIONS | |
| | | 13.3.1. | Sample Report | |
| | | 13.3.2. | I I | |
| | | 13.3.3. | General Analysis Conventions | 115 |

# 205801 | Statistical Analysis Plan RAP 08 Mar 2021 | TMF-1714066 | 3.0

# CONFIDENTIAL

| | | | 205801 |
|-------|---------|---------------------------------------------|--------|
| | 13.3.4. | Graphical Conventions | 115 |
| | 13.3.5. | P-values | 116 |
| | 13.3.6. | Use of Listings when Data Are Limited | 116 |
| | 13.3.7. | Considerations for Analysis of Interim Data | 116 |
| 13.4. | | SED DETAILED TABLE OF CONTENTS | |
| | 13.4.1. | Accrual and Study Status | 117 |
| | 13.4.2. | Baseline Characteristics | 117 |
| | 13.4.3. | Adverse Events | 118 |
| | 13.4.4. | Central Laboratory Measures | 118 |
| | 13.4.5. | Other Follow-up Measures | 119 |
| | 13.4.6. | Efficacy and Interim Analyses | 119 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology | <i>y</i> : | |
|---|---|---|
| 2017N337080_00 | 23-JUL-2018 | Original |
| 2017N337080_01 | 20-SEP-2018 | Amendment No.1 Protocol was amended at the request of the regulatory authority to provide additional clarification and guidance on specific aspects of the protocol |
| 2017N337080_02 | 15-JUL-2019 | Amendment No.2 Protocol was amended based on regulatory and ethics committee feedback to provide additional clarification and guidance on specific aspects of the protocol as described in the table in the protocol |
| 2017N337080_03 | 29-OCT-2020 | Amendment No.3 . Protocol was amended to add new substudies |
| TMF-11698443 | 02-FEB-2021 | Amendment No. 4. Protocol was amended to change the primary analysis criteria. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 4 (Dated: 02/FEB/2021).

# 2.2. Study Objective(s) and Endpoint(s)

# Part 1:

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| <ul> <li>To determine the safety and</li> </ul> | <ul> <li>AEs, SAEs, DLTs, changes in safety/laboratory</li> </ul> |
| tolerability of novel regimens | assessment parameters, dose modifications |
| Secondary Objectives | Secondary Endpoints |
| To provide a preliminary evaluation | Objective Response Rate (ORR) |
| of the efficacy of feladilimab in | Disease Control Rate (DCR) |
| combination with novel regimens | |
| Characterize the pharmacokinetic | PK parameters that include Cmax and Cmin for |
| properties of feladilimab (ICOS | feladilimab and in combination (and investigational |
| Agonist) or investigational | agent/s included in other arms), as data permit. |
| feladilimab combination partners | · · · |

205801

| Objectives | Endpoints |
|------------------------|-----------------------|
| Exploratory Objectives | Exploratory Endpoints |
| CCI | |

# Part 2:

| <ul> <li>Primary Objectives</li> <li>Determine whether experimental regimens provide evidence for improved survival over SoC therapy</li> <li>Evaluate milestone survival in participants treated with experimental regimens versus SoC therapy for NSCLC</li> <li>Evaluate other measures of antitumor activity of the experimental regimens compared with SoC therapy for NSCLC (RECIST 1.1 and iRECIST)</li> <li>Evaluate the safety and tolerability of the experimental regimens compared with SoC therapy for NSCLC</li> <li>Characterize the pharmacokinetic properties of feladilimab /SoC, or investigational feladilimab /soc densination partners</li> <li>Determine immunogenicity of experimental regimens</li> <li>Determine immunogenicity of experimental regimental regimens</li> <li>Determine immunogenicity of experimental regimental regimental regimental regimental regimental regim</li></ul> | Objectives | Endpoints |
|---|---|---|
| regimens provide evidence for improved survival over SoC therapy Secondary Objectives Evaluate milestone survival in participants treated with experimental regimens versus SoC therapy for NSCLC Evaluate other measures of antitumor activity of the experimental regimens compared with SoC therapy for NSCLC (RECIST 1.1 and iRECIST) Evaluate the safety and tolerability of the experimental regimens compared with SoC therapy for NSCLC (RECIST 1.2 and iRECIST) Frequency and severity of AEs, AESI; SAEs and AE/SAEs leading to dose modifications/delays/withdrawals; changes in laboratory, vital signs, and safety assessment parameters, including immunogenicity (ADA) Characterize the pharmacokinetic properties of feladilimab /SoC, or investigational feladilimab combination partners Determine immunogenicity of randomization to death milestone survival rate at 12 and 18 months Milestone survival rate at 12 and 18 months Milestone survival rate at 12 and 18 months PK, PR, SD, PD, PFS, ORR, DOR, DCR iCR, iPR, iUPD, iCPD, iSD iPFS; iORR; iDOR Frequency and severity of AEs, AESI; SAEs and AE/SAEs leading to dose modifications/delays/withdrawals; changes in laboratory, vital signs, and safety assessment parameters, including immunogenicity (ADA) PK parameters that may include Cmax and Cmin for feladilimab and SoC in combination (and investigational agent/s included in other arms) and for SoC alone, as data permit. | Primary Objectives | Primary Endpoints |
| <ul> <li>Evaluate milestone survival in participants treated with experimental regimens versus SoC therapy for NSCLC</li> <li>Evaluate other measures of antitumor activity of the experimental regimens compared with SoC therapy for NSCLC (RECIST 1.1 and iRECIST)</li> <li>Evaluate the safety and tolerability of the experimental regimens compared with SoC therapy for NSCLC</li> <li>Evaluate the safety and tolerability of the experimental regimens compared with SoC therapy for NSCLC</li> <li>Evaluate the pharmacokinetic properties of feladilimab /SoC, or investigational feladilimab combination partners</li> <li>Determine immunogenicity of</li> <li>Milestone survival rate at 12 and 18 months</li> </ul> | regimens provide evidence for improved survival over SoC | • |
| participants treated with experimental regimens versus SoC therapy for NSCLC Evaluate other measures of antitumor activity of the experimental regimens compared with SoC therapy for NSCLC (RECIST 1.1 and iRECIST) Evaluate the safety and tolerability of the experimental regimens compared with SoC therapy for NSCLC Characterize the pharmacokinetic properties of feladilimab /SoC, or investigational feladilimab combination partners CR, PR, SD, PD, PFS, ORR, DOR, DCR iCR, iPR, iUPD, iCPD, iSD iPFS; iORR; iDOR Frequency and severity of AEs, AESI; SAEs and AE/SAEs leading to dose modifications/delays/withdrawals; changes in laboratory, vital signs, and safety assessment parameters, including immunogenicity (ADA) PK parameters that may include Cmax and Cmin for feladilimab and SoC in combination (and investigational agent/s included in other arms) and for SoC alone, as data permit ADA incidence for feladilimab and combination | Secondary Objectives | |
| antitumor activity of the experimental regimens compared with SoC therapy for NSCLC (RECIST 1.1 and iRECIST) • Evaluate the safety and tolerability of the experimental regimens compared with SoC therapy for NSCLC • Characterize the pharmacokinetic properties of feladilimab /SoC, or investigational feladilimab combination partners • Determine immunogenicity of iCR, iPR, iUPD, iCPD, iSD iPFS; iORR; iDOR • Frequency and severity of AEs, AESI; SAEs and AE/SAEs leading to dose modifications/delays/withdrawals; changes in laboratory, vital signs, and safety assessment parameters, including immunogenicity (ADA) • PK parameters that may include Cmax and Cmin for feladilimab and SoC in combination (and investigational agent/s included in other arms) and for SoC alone, as data permit • ADA incidence for feladilimab and combination | participants treated with experimental regimens versus SoC | Milestone survival rate at 12 and 18 months |
| of the experimental regimens compared with SoC therapy for NSCLC NSCLC Characterize the pharmacokinetic properties of feladilimab combination partners Determine immunogenicity of AE/SAEs leading to dose modifications/delays/withdrawals; changes in laboratory, vital signs, and safety assessment parameters, including immunogenicity (ADA) PK parameters that may include Cmax and Cmin for feladilimab and SoC in combination (and investigational agent/s included in other arms) and for SoC alone, as data permit ADA incidence for feladilimab and combination | antitumor activity of the experimental regimens compared with SoC therapy for NSCLC | iCR, iPR, iUPD, iCPD, iSD |
| properties of feladilimab /SoC, or investigational feladilimab combination partners feladilimab and SoC in combination (and investigational agent/s included in other arms) and for SoC alone, as data permit • Determine immunogenicity of • ADA incidence for feladilimab and combination | of the experimental regimens compared with SoC therapy for | AE/SAEs leading to dose modifications/delays/withdrawals; changes in laboratory, vital signs, and safety assessment |
| | properties of feladilimab /SoC, or investigational feladilimab | feladilimab and SoC in combination (and investigational agent/s included in other arms) and |
| | experimental regimens | partners (where appropriate) |
| Exploratory Objectives Exploratory Endpoints | | Exploratory Endpoints |

205801



**Note**: The prefix "i", used for response related abbreviations in the above table indicates immune responses assigned using iRECIST.

# 2.3. Study Design



Between 10-20% of newly enrolled participants in subsequent substudies (depending upon the number of experimental arms in the trial) will be randomized to SoC once the initial 35 participants have been enrolled on control.

ICOS: Inducible T-Cell Co-Stimulator; NSCLC: non-small cell lung cancer; PD(L)1: Programmed Cell Death Protein 1 or Programmed Cell Death Ligand 1.

**Note:** Randomization of participants to experimental treatment regimens/arms may not occur in parallel. It should also be noted that the terms 'regimen' and 'arm' may be used interchangeably throughout the document.

# Design Features

- A randomized, open-label, platform trial utilizing a master protocol
- The study is structured as a series of substudies that share a common control arm
- The study has 2 parts, i.e. part 1 and part 2.
- Part 1 is a non-randomized part based on safety and pharmacokinetics/pharmacodynamics (PK/PD) evaluation.
- Part 2 is a randomized, Phase II part comparing the efficacy and safety of these novel regimens with SoC.
- Sub-study 1 has only part 2 and subsequent sub-studies (sub-studies 2,3 and 4) have both part 1 and 2
- Additional regimens may be added based on emerging nonclinical and clinical data, via future protocol amendment(s). This RAP will be upated as new arms are added.
- The study will evaluate the efficacy of feladilimab (ICOS Agonist) in combination with other treatment regimens compared with SoC (docetaxel) alone as the standard subsequent line chemotherapy Within Part 2 of each sub-study, patients will be randomized to receive either SoC or the experimental treatment; the randomisation ratios may change depending on the number of sub-studies running in parallel.
- Additional treatment arms may be added as sub-studies via future protocol amendments, and ongoing treatment arms may be dropped based on interim OS results or emerging safety information

205801

| Overview of St | udy Design a | and Key Fe | eatures | | | |
|---|---|---|---|---|---|---|
| Dosing | _ | - <u>-</u> | | T | T = - | |
| | | Sub- | Treatment | Dosage | Route of | Dosing |
| | 0 | <b>study</b><br>oC | Arm<br>Docetaxel | 75 | Administration IV infusion | Frequency<br>Once Q3W |
| | 0 | 00 | Docetaxei | mg/m <sup>2</sup> | TV IIIIUSIOII | Office QSW |
| | S | ub-study | feladilimab | 80 mg | IV infusion | Once Q3W |
| | 1 | | Docetaxel | 75<br>mg/m <sup>2</sup> | IV infusion | Once Q3W |
| | S<br>2 | ub-study | Ipilimumab | 1 mg/kg | IV infusion | Once Q3W |
| | | | | 3 mg/kg | | |
| | | | feladilimab | 24mg | IV infusion | Once Q3W |
| | S<br> 3 | ub-study | Niraparib | 200 mg <sup>a</sup><br>300 mg <sup>b</sup> | Oral | Daily |
| | | | feladilimab | 24mg | IV infusion | Once Q3W |
| | | ub-study | Dostarlimab | 500 mg | IV infusion | Once Q3W |
| | 4 | | Cobolimab | 300 mg | IV infusion | Once Q3W |
| | | | feladilimab | 24mg | IV infusion 77 kg or baseline plate | Once Q3W |
| Time & | ≥18 Ex the pro def def Sir dea | b: For participants with baseline body weight ≥77 kg and baseline platelet count ≥150,000/µL. Experimental treatment (combination) will continue to be administered at the indicated schedule with the maximum duration as specified in the protocol for each combination arm, or until disease progression as determined by iRECIST, death, unacceptable toxicity, or other protocoldefined criteria are met. Single agent SoC treatment may continue until disease progression, death, unacceptable toxicity, withdrawal of consent, or per insitiutional standard for docetaxel. | | | | |
| Events | - | | ix 2: Schedule | | | |
| Treatment<br>Assignment | subsequent sub-studies (depending upon the number of experimental arms in the trial) will be randomized to SoC once the initial 35 participants have been enrolled on control. Once determined to be eligible for the study, all participants will be centrally randomized using RAMOS, an Interactive Web Response System (IWRS). | | | | | |
| Interim<br>Analysis | <ul> <li>No interim analysis is involved in part 1</li> <li>In part 2, interim analyses focusing on safety (also including OS) will be performed approximately every 3 to 6 months depending on the amount of additional data accrued. These interims would be conducted across all substudies, reported by treatment and SoC will be combined across all substudies.</li> </ul> | | | | | |

#### **Overview of Study Design and Key Features**

- An interim analysis of OS will be conducted for each experimental arm after approximately 45 events (experimental arm and SoC combined) and a minimum of 18 events from experimental arm have been observed.
- Interim analysis will assess futility. Success will only be declared at the final analysis.
- Interim analysis will be performed by an independent third party Statistical Data Analysis Center (SDAC) and details of Interim Analysis Plan will not be described in this document but will be described in SDAC Reporting Plan (Section 12.12)

# 2.4. Statistical Hypotheses / Statistical Analyses

# 2.4.1. Hypothesis

**Part 1:** The primary objective of Part 1 is to establish the safety and tolerability of the experimental combination regimen of each substudy.

#### Part 2:

The primary objective of the study is to determine whether the experimental arms prolong overall survival relative to standard of care (SoC).

The null hypothesis is that there is no difference in overall survival between each experimental arm and the SoC and alternative hypothesis is that the experimental regimen improves overall survival over the SoC. No comparisons will be made between experimental arms.

The predictive probability inference approach will be used as the basis for both interim and final success decision making. The predictive probability of Phase III study success (defined as a statistically significant log-rank test with1-sided alpha=0.025) will be calculated as a measure of the improvement in OS in the experimental arm compared with the SoC arm.

As this is a signal finding study and not confirmatory, each experimental arm will be compared to control in a pairwise fashion with no adjustment for multiple comparisons.

#### 2.4.2. Sample Size

#### Part 1:

A maximum of 15 participants will be enrolled to each scheduled regiment in Part 1.

#### Part 2:

In Part 2, 70 participants in each experimental arm and a minimum of 35 participantes in the SoC arm will be randomized. Sample size and associated operating characteristics were evaluated via simulation.

205801

The 8-month milestone survival in the SoC arm is estimated to be  $\sim$ 40% in advanced squamous cell lung cancer (Brahmer, 2015),  $\sim$ 60% in advanced non-squamous lung cancer (Borghaei, 2015), and  $\sim$ 50% in PD-L1 positive population (Herbst, 2016). The participant population in the current study is expected to be a mixed population with both squamous and nonsquamous lung cancer participants; therefore, mean target rate is assumed to be  $\sim$ 50% (Figure 1).

For the target effect of experimental regimens, there is a potential delayed effect at treatment start and sustained effect after prolonged follow-up (Brahmer, 2015; Borghaei, 2015). The survival probability in these arms is expected to overlap that in the SoC arm for up to 4 months from start of treatment followed by a separation. It is hypothesized that percentage of surviving participants is maintained at 20% after 24 months (Figure 1).

Under the alternative hypothesis, three-piece piecewise Weibull distributions are used to describe the survival distribution of each experimental arm and two-piece piecewise Weibull distributions are used to describe the survival curve of docetaxel (Table 48 in Section 12.13.1 of the protocol describes the simulation parameters). Using this modelling approach for the primary endpoint of OS, the assumed survival curve for the SoC arm is presented using blue dashes and the target survival curve for the experimental arm is presented as the solid red curve in Figure 1. Based on these two curves, the hazard ratio is approximately 0.58.

Sample size was chosen by simulating the a study in which 4 experimental arms enter the master protocol at different points in time. Enrollment of 9 participants per month is assumed. Interim and final analyses are performed based on predetermined decision rules as specified in Section 3. The planned Phase III sample size is 300 (150 participants per arm and a total of 210 events). The future phase 3 trial will use the log-rank (frequentist) test and the decision rule at interim and end of phase 2 will use the (Bayesian) predictive probability, given the results in phase 2, that the future log-rank test in phase 3 will be significant, thus, resulting in a methodology that is a mixture of Bayesian and frequentist. Simulations assess the Operating Characteristics of the predictive probability decision criteria under the null and alternative hypotheses. A cutoff of 43% or greater for the predictive probability of phase 3 success is used to define success for each experimental arm. Sample size was calculated under the simulated survival curves shown below (Figure 1).

The final analysis of OS for a substudy will be performed when approximately 85 death events have occurred in the experimental arm and SoC arm combined, and the last participant in that substudy has been randomized for at least 6 months. In the case death events occur at a rate lower than expected due to potentially prolonged survival benefit, to avoid substantial delay of final analysis for a substudy, the primary analysis for a substudy may be conducted once approximately 75 events have occurred and the last participant in that substudy has been randomized for at least 6 months, at the discretion of the Sponsor. A minimum of 35 events are needed from the experimental arm for both primary and final analysis.

Assuming the true HR $\approx$ 0.58, 85 death events will provide 94.2% probability (power) of achieving the predictive probability success criteria for future phase 3 success of  $\geq$  43%.

In the case of primary analysis being performed with 75 death events, it will provide 88.3% probability of achieving the predictive probability success criteria. If the true HR is 1, 85 and 75 death events will provide 16.6% and 18.2% probability of achieving the predictive probability success criteria (Type I error), respectively

Figure 1 Assumed Survival Probability Under Alternative Hypothesis in Experimental Regimnes (Red) and Docetaxel (Blue)



# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

#### Part 1:

No interim analysis will be performed in part 1 of the study

#### Part 2:

This is a platform study utilizing a master protocol designed so that experimental arms may enter and leave the trial independently at different time points as determined by prespecified decision criteria. This study will be conducted under the auspices of an IDMC and Steering Committee. The IDMC will review all available interim safety and efficacy (OS only) data as the study progresses. The details of the data that will be reviewed by IDMC is described in the IDMC charter and/or the SDAC Reporting Plan (Section 12.12). The Steering Committee will provide guidance over key decision points during the conduct of the study including, but not limited to, the introduction of new experimental arms into the master protocol, graduation of existing arms for further development in other studies, and end of study. The SoC may be changed during the course of the study and this may require update to the RAP and study protocol.

Interim analyses will be performed approximately every 3 to 6 months depending on the amount of additional data accrued.

For each experimental arm, an interim analysis of OS will be performed. The study may be stopped for futility at this interim analysis.

#### 3.1.1. Interim Analyses for Overall Survival (OS)

Interim Analysis will be performed by Statistical Data Analysis Center (SDAC) for IDMC.

OS is defined as the interval from date of randomization to the date of death, irrespective of the cause of death. If a participant does not have a documented date of death or is lost to follow-up, time of death will be censored at the date of last contact.

An interim analysis of OS will be conducted for each experimental arm after approximately 45 events (experimental arm and SoC combined) and a minimum of 18 events from experimental arm have been observed. Interim analyses will not be used to declare success of any experimental arm.

The study will employ a Bayesian decision-making framework based on the predictive probability of observing a significant improvement in OS in a future Phase III trial. The predictive probability inference approach will be used as the basis for interim analyses. The predictive probability of Phase III study success (defined as a statistically significant improvement in OS, 1-sided alpha=0.025) will be calculated as a measure of the improvement in OS in the experimental arm compared with the SoC arm. Each experimental arm will be compared to the SOC arm in a pairwise fashion with no adjustment for multiple comparisons.

If the predictive probability of phase 3 success for a particular experimental arm is very low (as defined in the IDMC charter and/or SDAC Reporting Plan (Section 12.12), that experimental arm may be considered for termination. Final decision on termination of an experimental arm will be based on the totality of the data, which will include the calculated predictive probability of success and the available safety data for that experimental arm.

# 3.2. Primary and Final Analyses

The final planned primary analyses for each experimental arm will be performed after the completion of the following sequential steps:

#### Part 1:

- 1. A futility analysis of ORR will be conducted after 10 participants have had at least two post baseline RECIST assessments.
- All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. Randomization codes have been distributed according to RandAll NG.

#### Part 2:

- 1. The final analysis for each experimental arm will occur after observing approximately 85 events (experimental regimen and SoC combined) with minimum of 35 events in the experimental arm.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. Randomization codes have been distributed according to RandAll NG.

The rest of the data on remaining subjects will be reported appropriately at study end. The RAP will be updated accordingly for each sub study.

In the case death events occur at a rate slower than expected due to potentially prolonged survival benefit, to avoid substantial delay of final analysis for a substudy, primary analysis for a substudy may be conducted once approximately 75 events have occurred and at least 35 events observed in the experimental arm, and the last participant in that substudy has been randomized for at least 6 months, at the discretion of the Sponsor.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility. | <ul> <li>Study Population</li> </ul> |
| Safety | All randomized participants who received at least one dose of SoC or experimental regimen based on actual treatment received. | Safety |
| Intent-To-Treat<br>(ITT) | All participants who were randomized to treatment<br>regardless of whether the participants actually<br>received study treatment. | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Pharmacokinetic (PK) | All participants in the safety population from whom at least one blood sample was obtained and analysed for PK concentration. | PK Concentration<br>and PK<br>parameters |
| DLT Evaluable | <ul> <li>A subset of participants in part 1 who have received the first course of treatment containing both agents within a sub-study and followed up for a 21-day period or withdrawn within 21 days due to an AE meeting the definition of a DLT.</li> <li>For oral dosing, a participant is considered DLT evaluable if they received at least 80% the first course of treatment containing both agents within a sub-study and followed up for a 21-day period or withdrawn within 21 days due to an AE meeting the definition of a DLT</li> </ul> | • DLT |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important and non-important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and important protocol deviations will be listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reporting | |
| Code | Description | Description | Order in TFL |
| S | Standard of Care Docetaxel 75 mg/m2 | Docetaxel | 1 |
| A | GSK3359609 (ICOS Agonist)<br>80 mg plus docetaxel<br>(Treatment Regimen 1) | GSK3359609 80 mg<br>plus Docetaxel 75<br>mg/m2 | 2 |
| Е | GSK3359609 (ICOS Agonist)<br>plus 1 mg/kg Ipilimumab<br>(Treatment Regimen 2) | Feladilimab 24 mg plus<br>Ipilimumab 1 mg/kg | 2 |
| F | GSK3359609 (ICOS Agonist)<br>plus 3 mg/kg Ipilimumab<br>(Treatment Regimen 3) | Feladilimab 24 mg plus<br>Ipilimumab 3 mg/kg | 3 |
| G | GSK3359609 (ICOS Agonist)<br>plus Niraparib (Treatment<br>Regimen 4) | Feladilimab 24 mg plus<br>Niraparib | 2 |
| Н | GSK3359609 (ICOS Agonist)<br>plus Dostarlimab plus<br>Cobolimab (Treatment<br>Regimen 5) | Feladilimab 24 mg plus<br>Dostarlimab 500 mg<br>plus Cobolimab 300 mg | 2 |

#### 5.2. Baseline Definitions

- For all endpoints the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. For laboratory data, baseline will be the latest non-missing pre-dose value from local lab will be used.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Multicentre Studies

In this multicentre and multi-country study, enrolment will be presented by country and investigative site. All centres will be pooled prior to analysis.

Additional displays on specific region may be explored as data warrants.

# 5.4. Examination of Covariates, Other Strata and Subgroups

#### Part 1:

No stratification and subgroup analysis is performed in part 1.

#### Part 2:

#### 5.4.1. Covariates and Other Strata

The list of covariate and strata described below may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses if data permits. Additional covariates and other strata of clinical interest may also be considered as data warrants.

| Category | Details |
|----------|------------------------------------|
| Strata | Squamous vs. Non-squamous |
| | Line of PD(L)1 therapy 1st vs. 2nd |

# 5.4.2. Examination of Subgroups

Subgroups may be explored as the study progresses. Subgroup analysis may be performed if data permits. In addition to the strata listed above, subgroups of interest may include Gender and Age.

| Subgroup | Categories |
|----------|--------------|
| Gender | Male; Female |
| Age | <65; ≥65 |

# 5.5. Multiple Comparisons and Multiplicity

Each experimental arm will be compared to control in a pairwise fashion with no adjustment for multiple comparisons. No formal comparisons will be made between experimental arms.

205801

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the ITT, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, past and current medical conditions, prior and concomitant medications, disease characteristics at initial diagnosis and at screening, prior and follow-up anti-cancer therapy, surgical/medical procedures, substance use, duration of follow up, will be based on GSK Core and Oncology Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

# 6.2. Disposition of Subjects

A summary of the number of subjects in each of the analysis populations described in Section 4 will be provided. Number of subjects based on the ITT will be summarized by country and site for each cohort.

A summary of subject status and reason for study withdrawal will be provided. This display will show the number and percentage of subjects who have completed the study or have withdrawn from the study, including primary and secondary (if any) reasons for study withdrawal. Reasons for study withdrawal will be presented in the order they are displayed in the eCRF (Electronic Case Report Form). Subjects who die for any reason during on-treatment period will be considered to have completed the study.

A summary of study treatment status will be provided. This display will show the number and percentage of subjects who discontinued study treatment and a summary of the primary reasons for discontinuation of study treatment. Reasons for study treatment discontinuation will be presented in the order they are displayed in the eCRF.

A listing of treatment discontinuation will be generated. The listing will include last dose date and primary reasons for study treatment discontinuation.

The number and percentage of subjects who passed screening and entered the study, who failed screening and therefore were not entered into the study, and subjects who met eligibility criteria but were not needed will be summarized along with the reasons for failure will be summarized for those subjects who failed screening. A subject may have more than one reason for screen failure.

Since screen failures are not assigned to treatment groups, the display has only one subject-group column regardless of study design. Also, since screen failures cannot be attributed to any of the sub-studies repeat reporting may occur in different sub-studies/parts. This summary will be based on the Screened population.

The number of subjects will be summarized by Country, Site ID and Investigator ID. This summary must be produced based on the all enrolled population. The total column, summarizing subjects regardless of treatment, should always be included. Rows should be sorted alphabetically by country, then in numerical order by Site ID

# 6.3. Demographic and Baseline Characteristics

The demographic characteristics (e.g., age, race, ethnicity, sex, height, and baseline body weight) will be listed and summarized. Age, height and weight will be summarized using the mean, standard deviation, minimum, median, and maximum. In addition, age will also be categorized and summarized by 18-64, 65-74, 75-84, and ≥85. The count and percentage will be computed for race, ethnicity and sex.

A separate summary of age ranges based on the ITT population will be provided. Age will be summarized in categories: 18-64, 65-84, and ≥85. Race and racial combinations will also be summarized. Listing of Race will also be provided.

#### 6.4. Prior Medical Condition and Disease Characteristics

Disease history and characteristics (primary tumor type, lesion status, time since initial diagnosis, stage at initial diagnosis, time since last progression) will be summarized. Indicators (yes/no) for the following, collected at screening, will also be summarized: measurable disease, non-target lesions, and metastatic disease. Medical conditions present at screening will be listed and will be summarized by past and current. Disease history and characteristics, as well as these medical conditions, will be presented in data listings.

A summary of disease burden at baseline will be provided. Information on sites of metastatic disease at screening will be summarized.

Prior cancer related surgeries will be summarized and listed.

# 6.5. Prior and Subsequent Anti-cancer Therapy

Anti-cancer therapy will be coded using GSK Drug dictionary version 1.6 or higher. Prior anti-cancer therapy will be coded using GSK Drug coding dictionary, then summarized by type of therapy and listed. A listing of prior anti-cancer therapy will show the relationship between Anatomical Therapeutic Chemical (ATC) Level 1, ingredient, and verbatim text; therapies will be classified by type (chemotherapy, immunotherapy, hormonal therapy, biologic therapy, radioactive therapy, small molecule targeted therapy, surgery and radiotherapy).

ATC classification Level 1 (Body System) information will be included in the dataset created but will not appear on the listing or summary.

The prior and follow-up anti-cancer therapies will be summarised by ingredient. The number and percentage of subjects that received different types of anti-cancer therapies ((chemotherapy, immunotherapy, hormonal therapy, biologic therapy, radioactive therapy, small molecule targeted therapy, surgery and radiotherapy) as prior therapy and

205801

follow-up therapy will be summarised separately. A subsequent listing of the type of Anti-cancer therapy received will be provided with an indicator variable(Yes/No) for Prior and Follow-up anti-cancer therapy and prior radio therapy

#### 6.6. Concomitant Medications

Prior medications will be coded using GSK Drug coding dictionary and summarized. The summary of prior medications will show the number and percentage of subjects taking prior medications by Ingredient.

Concomitant medications will be coded using GSK Drug coding dictionary and summarized. The summary of concomitant medications will show the number and percentage of subjects taking concomitant medications by Ingredient. Multi-ingredient products will be summarized by their separate ingredients rather than as a combination of ingredients.

In the summary of concomitant medications, each subject is counted once within each unique ingredient. For example, if a subject takes Amoxicillin on two separate occasions, the subject is counted only once under the ingredient "Amoxycillin". In the summary of concomitant medications, the ingredients will be summarized by the base only, using CMBASECD and CMBASE.

Concomitant medications will be summarized separately for medications with onset date within the on-therapy period and for medications with onset date within the pre-therapy period. Note: In order to be considered a concomitant medication, the concomitant medication must have been taken at some point during the on-therapy window.

Blood products or blood supportive care products with onset date within the on-therapy window will be included in the summary tables. The frequency and percentage of subjects using blood products and blood supportive care products after the start of study treatment will be provided. Supportive listings will also be provided.

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

# 7.1.1. Endpoint / Variables

There is no primary efficacy analysis or endpoint for Part 1.

The primary efficacy analyses for Part 2 will be based on the ITT population, unless otherwise specified and all summaries and data listings will use treatment labels as specified in Section 5.1.

Primary endpoint is OS and primary analysis is based on the predictive probability of Phase III study success.

**Overall Survival (OS)** is defined as the time from randomization to the date of death for any cause. In the absence of confirmation of death, survival time will be censored at the last date the subject is known to be alive (i.e., at their last known alive date from long term follow-up).

The length of OS will be calculated as

OS = death date or last known alive date - date of randomisation + 1

Subjects lacking data beyond date of randomisation will have their survival times censored at date of randomisation.

# 7.1.2. Summary Measure

Hazard Ratio for OS will be estimated using the cox proportional hazard model stratified by the histology(squamous vs. non-squamous) and line of PD-L1 therapy(1<sup>st</sup> line vs. 2<sup>nd</sup> line) with treatment arm as the sole explanatory variable.

The distribution of OS for each treatment arm will be estimated using the Kaplan-Meier method. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of OS will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method (Brookmeyer, 1982).

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the ITT population, unless otherwise specified.

#### 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# **Endpoint / Variables**

OS

#### **Model Specification**

- Hazard ratio for OS and corresponding 95% confidence interval will be estimated using the Cox's proportional hazard model stratified by stratified by the histology(squamous vs. non-squamous) and line of PD-L1 therapy(1st line vs. 2nd line) with treatment arm as the sole explanatory variable.
- The predictive probability of Phase III study success (defined as a statistically significant log-rank test with 1-sided alpha=0.025) will be calculated as a measure of the improvement in OS in the experimental arm compared with the SoC arm.
- The predictive probability of success in a future Phase III study will be calculated using the posterior predictive distribution of log(HR in phase 3), given log(HR from phase 2), assuming that both the observed log(HR) and prior for mean of log(HR) follow normal distributions as outlined below.
- Let us assume that the prior of hazard ratio (in logarithm scale) follows normal distribution with mean as  $\theta_0$  and a standard deviation of sqrt(4/n<sub>0</sub>)

$$\theta \sim N(\theta_0, V_0)$$

where  $V_0 \sim 4/n_0$ ,  $n_0$  = some number that could be interpreted as the number of events in a trial where the prior information came from; a small value corresponds to a large variance for the prior distribution and thus, the prior is considered non-informative. The expression for the variance comes from (Parmar, 1998) if the trial where the prior info was obtained has equal sample size allocation between the 2 groups.

• The posterior distribution is also normal (Gelman, 2013) and is given by:

$$\theta | x \sim N \left( \frac{V_0}{V_{p2} + V_0} x + \frac{V_{p2}}{V_{p2} + V_0} \theta_0, \frac{1}{1/V_0 + 1/V_{p2}} \right).$$

• The *posterior* predictive distribution, given the observed data in phase 2, is normal (Gelman, 2013) and is of the form

$$y|(X=x) \sim N\left(\frac{V_0}{V_{p2} + V_0}x + \frac{V_{p2}}{V_{p2} + V_0}\theta_0, \frac{1}{1/V_0 + 1/V_{p2}} + V_{p3}\right)$$

where 
$$V_{p3} = V[\log(\widehat{HR}_{p3})]$$

• and  $V_{p3}$  is assumed to be known. If the numerator and denominator of the expression for the mean is divided by  $(V_0V_{p2})$ , the posterior predictive distribution is of the form

$$Y|x \sim N \left( \frac{\frac{V_0}{V_0 V_{p2}}}{\frac{V_{p2}}{V_0 V_{p2}} + \frac{V_0}{V_0 V_{p2}}} x + \frac{\frac{V_{p2}}{V_0 V_{p2}}}{\frac{V_{p2}}{V_0 V_{p2}} + \frac{V_0}{V_0 V_{p2}}} \theta_0, \frac{1}{1/V_0 + 1/V_{p2}} + V_{p3} \right)$$

and could be expressed as

$$Y|x \sim N \left( \frac{\frac{1}{V_{p2}}}{\frac{1}{V_0} + \frac{1}{V_{n2}}} x + \frac{\frac{1}{V_0}}{\frac{1}{V_0} + \frac{1}{V_{n2}}} \theta_0, \frac{1}{1/V_0 + 1/V_{p2}} + V_{p3} \right)$$

or equivalently

$$Y|x \sim N \left( \frac{\frac{x}{V_{p2}} + \frac{\theta_0}{V_0}}{\frac{1}{V_0} + \frac{1}{V_{p2}}}, \frac{1}{1/V_0 + 1/V_{p2}} + V_{p3} \right).$$

• The planned future phase 3 trial will have equal sample size allocation for the 2 groups and the total number of events in this phase 3 trial is m. We also assume that  $V_{p3}$  is known with value given by its estimate from (Parmar, 1998)

$$V_{p3} \approx \frac{4}{m}$$
.

• The predictive posterior distribution, with  $V_{p3}$  replaced by its estimate, is of the form given in protocol Section 10.5.1 and as shown below

$$Y|x \sim N \left(\frac{\frac{x}{V_{p2}} + \frac{\theta_0}{V_0}}{\frac{1}{V_0} + \frac{1}{V_{p2}}}, \frac{1}{1/V_0 + 1/V_{p2}} + \frac{4}{m}\right).$$

• If we assume that the prior distribution is non-informative such that  $V_0$  is a very large number relative to  $V_{p2}$ , then the posterior predictive distribution (Gelman, 2013) is given could be reduced to

$$Y|x \approx N(x, V_{n2} + V_{n3}).$$

• Success in future phase 3 is defined as "observing a statistically significant one-sided 2.5% alpha-level log-rank test in a trial where sample size allocation in 2 groups is equal and the total number of events in the trial is m." The log-rank test statistic in the future phase 3 trial could be expressed as

$$Z_{p3} = \left(\log(\widehat{HR}_{p3}) * \sqrt{\frac{m}{4}}\right) \approx N(0,1).$$

• Under the null hypothesis of equality of hazard in phase 3, the one-sided 2.5% alpha-level log-rank test is statistically significant if

$$Z_{p3} < -1.96$$
 or equivalently,  $y = \log(\widehat{HR}_{p3}) < -1.96 * \sqrt{\frac{4}{m}}$ .

- The probability of phase 3 success given phase 2 data is calculated using the predictive distribution of Y given X=x. This is the area under the posterior predictive distribution of Y given X=x in the region  $Y < -1.96 * \sqrt{4/m}$ , by virtue of the additional assumption that  $V_{p2}$  and  $V_{p3}$  are known. If  $\Phi(\cdot)$  denotes the standard normal distribution function (i.e.,  $\Phi(-Z_{\alpha}) = \alpha$ ), then the predictive probability of phase 3 success, given phase 2 data, is calculated as
- $\bullet \quad \Phi \left( \frac{-1.96*\sqrt{\frac{4}{m}} \left(\frac{\frac{x}{V_{p2}} + \frac{\theta_0}{V_0}}{\frac{1}{V_0} + \frac{1}{V_{p2}}}\right)}{\sqrt{\frac{1}{\sqrt{V_0} + \frac{1}{V_{p2}}} + \frac{4}{m}}} \right).$
- Assuming Non-informtaitve Prior, i.,e.  $V_0$  is very large [relative to  $V_{p2}$

$$Y|x \sim N \left( \left[ \frac{V_0}{V_{p2} + V_{p0}} \right] x + \left[ \frac{V_2}{V_2 + V_0} \right] \theta_0, \left( \frac{1}{\left[ \frac{1}{V_0} \right]} + \left[ \frac{1}{V_{p2}} \right] + V_3 \right) \right)$$

$$Y|x \sim N \left( \left[ \frac{V_0}{V_{p2} + V_{p0}} \right]^{\frac{1}{2}} x + \left[ \frac{V_2}{V_2 + V_0} \right]^{\frac{0}{2}} \theta_0, \left( \frac{1}{\left[ \frac{1}{V_0} \right]^{\frac{0}{2}} + \left[ \frac{1}{V_{p2}} \right]} + V_3 \right) \right)$$

$$Y|x \approx N \left( x, \left( V_{p2} + V_3 \right) \right)$$

• Therefore, Phase 3 PoS given Phase 2 Data is:

$$P(Y < -1.96\sqrt{V_3} \mid x)$$

This is area under Posterior Predictive Distribution of

$$Y|x \sim N\left(x, \left(V_{p2} + V_3\right)\right)$$

• Equivalently, this is the area under N(0,1) to the left of

$$V[log(sample\ HR)] = \left(\frac{\frac{(-1.96\sqrt{V_3}) - x}{\sqrt{V_{p_2} + V_3}}}{\frac{1}{\sqrt{V_{p_2} + V_3}}}\right) + \left(\frac{1}{\#\ Events\ in\ Treatment}\right)$$

Therefore:

$$V_{p2} = V[log(sample\ HR)\ from\ phase\ 2] \approx \frac{1}{n_c} + \frac{1}{n_t}$$
  
 $V_3 = V[log(sample\ HR)\ in\ phase\ 3] \approx \frac{4}{m}$   
note: m = total # events in a 2-arm study with equal allocation

• At final analysis, PoS is area under N(0,1) to the left of

$$\frac{\left(-1.96\sqrt{V_3}\right)-x}{\sqrt{V_{n2}+V_3}}$$

or equivalently

$$\frac{\left(-1.96\sqrt{\frac{4}{m}}\right) - log(sample HR from platform trial)}{\sqrt{\frac{1}{n_c} + \frac{1}{n_t} + \frac{4}{m}}}$$

# **Model Checking & Diagnostics**

- Before using the cox proportional hazard model, the proportional hazards assumption will be assessed using the following methods:
  - Kaplan-Meier plot by treatment arm
  - Plot of log(time) against log(-log(survival)) by treatment arm
  - Plot of Schoenfeld residuals for treatment
  - Evaluation of time-dependency of treatment effect by adding an interaction term of treatment and time in the Cox model. If the interaction term is significant (p< 0.05), it is considered that the proportional hazards assumption is violated.
- If one or more of the tests above demonstrates clear violation of the proportional hazards assumption, it is considered the proportional hazards assumption does not hold. Hazard ratio and corresponding 95% CI estimated from the Cox model will still be reported.

#### **Model Results Presentation**

 Cox proportional hazard model results will be summarised in tables accounting for the stratification factors. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of OS will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method (Brookmeyer, 1982) and presented in tables. In addition Kaplan Mier figures will presented to show the distribution of OS.

# Sensitivity and Supportive Analyses

 If the proportional hazard assumption does not hold, additional analysis based on (Restricted Mean Survival Time) RMST may be explored.

205801

- Sensitivity analyses will be conducted to evaluate time-dependency in the SoC arm. The exchangeability assumption will be examined by comparing overall survival between non-concurrent and concurrent SoC data, by using Cox's proportional hazard model with indicator in control data (0: nonconcurrent, 1: concurrent data) as a covariate. If there is a difference in OS between non-concurrent and concurrent SoC, this difference will be further investigated or examined. Sensitivity analysis will be conducted if there is evidence of a violation of the exchangeability assumption. An example of a sensitivity analysis is one where only the concurrent data will be included (i.e., no non-concurrent data are used) in evaluating the treatment effect of the experimental regimen at data analysis.
- A sensitivity analysis may be performed to adjust for the impact of COVID 19. The censoring rule as described below will be followed.
  - a. Participants will be censored at the earliest date of,
    - Treatment discontinuation related to COVID -19 and not associated with disease progression
    - Death due to COVID-19 infection and not associated with disease under study
  - b. If none of the above events (i & ii) occurs and an event death occurs, the event will be based on the date of death due to any cause other than COVID-19 infection.
  - c. Else if both a and b didn't occur then the participants will be censored at last known alive date, as per the primary analysis censoring rules.

# 7.2. Secondary Efficacy Analyses

#### 7.2.1. Endpoint / Variables

#### **Part 1:**

The secondary efficacy analyses for Part 1 will be based on safety population unless otherwise specified. The secondary endpoints in part 1 are, Overall Response Rate (ORR) and Disease Control Rate (DCR).

**ORR** is defined as the percentage of participants with a best overall confirmed CR or PR at any time as per RECIST1.1

**DCR** is defined as the percentage of participants with best overall confirmed complete response, partial response or stable disease at any time as per RECIST1.1

Summary measures for ORR and DCR will be provided as mentioned in Section 7.2.3.

# Part 2:

The secondary efficacy analyses for Part 2 will be based on the ITT population, unless otherwise specified and all summaries and data listings will use treatment labels as specified in Section 5.1. The key secondary efficacy endpoint is Milestone Survival rate at 12 and 18 months. Other secondary endpoints are CR, PR,SD, PD, PFS, ORR, DOR, iCR, iPR, iUPD, iCPD, iSD, iPFS, iORR and iDOR which were used to evaluate anticancer activity.

- Milestone Survival rate at 12 months is defined as the percentage of people alive until 12 months after randomisation. It is the time from date of randomization to the date of death due to any cause during the period of 12 months. In the absence of confirmation of death during the period of 12 months, survival time will be censored at the last contact date. If the death date or date of last contact date is after 12 months then the censor date will be randomisation date + 12 months.
- Milestone Survival rate at 18 months is defined as the percentage of people alive until 18 months after randomisation. It is the time from date of randomization to the date of death due to any cause during the period of 18 months. In the absence of confirmation of death during the period of 18 months, survival time will be censored at the last contact date. If the death date or date of last contact date is after 18 months then the censor date will be randomisation date + 18 months.

The length of **Milestone Survival** will be calculated as

Milestone Survival = death date or last available date (during the period of 12 or 18 months) – date of randomization + 1

205801

Subjects lacking data beyond date of randomisation will have their survival times censored at date of randomisation

The **Milestone Survival Rate** will be calculated as the (Kaplan Meir survival probabilities at time points 12 months/18 months) \* 100.

For Anti-cancer activity Analyses, ITT population will be used unless otherwise specified. Anticancer activity will be evaluated based on clinical evidence and response criteria. The response data will be summarized by each treatment (iRECIST will be used for response endpoints and disease measurements for iORR, iDOR and iPFS; RECIST 1.1 guidelines will be used for response endpoints and disease measurements for ORR, DOR and PFS).

ORR, DCR, DOR and PFS as well as iORR, iDCR, iDOR and iPFS will be calculated and summarized.

**ORR or iORR** is defined as the percentage of participants with a best overall confirmed CR or PR at any time as per RECIST1.1/iRECIST.

**DCR or iDCR** is defined as the percentage of participants with best overall confirmed complete response, partial response or stable disease at any time as per RECIST1.1/iRECIST 1.1.

**Best overall response (BOR)** or **iBOR** will be derived on investigator assessments of oveall response at each visit recorded from the start of treatment until the criteria for progression are met (considering any requirement for confirmation when needed), or the date of initiation of new anti-cancer therapy (Note: This excludes palliative radiotherapy), or death date, whichever is earliest, as assessed by the investigator per RECIST 1.1 /iRECIST criteria.

For RECIST 1.1,

To be assigned a status of confirmed CR/PR, a confirmatory disease assessment should be performed no less than 4 weeks (28 days) after the criteria for response are first met.

Responses of CR/PR that do not meet the requirements of confirmed CR/PR are still eligible to be considered SD if it has met the SD criteria.

For RECIST 1.1, to be assigned a status of SD, follow-up disease assessment(s) must have met the SD criteria at least once after the first dose at a minimum of 8 weeks (56 days) from baseline. If the minimum of 8 weeks (56 days) for SD is not met, the best overall response will depend on the subsequent assessments. For example, if an assessment of PD follows the assessment of SD and SD does not meet the minimum 8-week requirement the best response will be PD. Alternatively, subjects lost to follow-up after an SD assessment not meeting the minimum time criteria will be considered not evaluable.

205801

For iRECIST, confirmatory disease assessment of PR or CR will be performed no less than 4 weeks (28 days) after the criteria for response are first met. In addition, a confirmatory disease assessment of PD will be performed no less than 4 weeks and up to 8 weeks later to confirm PD.

If NE (Not Evaluable) is recorded in between initial and confirmatory (i)CR or (i)PR or inbetween iUPD and iCPD then it can disregarded to obtain the Best Response

A SD in between an intial PR and confirmation PR can also be disregarded to obtain the Best Response of PR (see below table)

An iUPD between initial (i)CR/(i)PR and confirmed (i)CR/(i)PR can also be disregarded, as this can be considered to be a pseudo-progression

| Assessment<br>1 (overall<br>reponse) | Assessment 2 (overall reponse) | Assessment 3 (>= 4 weeks after) (overall reponse) | Assessment<br>4 (overall<br>reponse) | Best Response |
|---|---|---|---|---|
| (i)CR | NE | (i)CR | - | (i)CR |
| (i)PR | NE | (i)PR | - | (i)PR |
| (i)PR | SD | (i)PR | - | (i)PR |
| (i)CR | NE | NE | (i)CR | (i)CR |
| (i)PR | NE | NE | (i)PR | (i)PR |
| iUPD | NE | NE | iCPD | iCPD |
| (i)CR | iUPD | (i)CR | - | (i)CR |
| (i)PR | iUPD | (i)PR | - | (i)PR |
| (i)PR | iUPD | iUPD | (i)PR | (i)PR |

**DOR or iDOR** is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause among participants who achieve an overall response (i.e., unconfirmed or confirmed CR or PR). Censoring rules will follow those of the PFS analysis.

**PFS or iPFS** defined as time from the date of randomization to the date of disease progression per clinical or radiological assessment or death due to any cause, whichever occurs earlier. For the analysis of PFS, if the participant received subsequent anticancer therapy prior to the date of documented events, PFS will be censored at the last adequate assessment (e.g., assessment where visit level response is CR, PR or SD) prior to the initiation of therapy. Otherwise, if the participant does not have a documented date of event, PFS will be censored at the date of the last

adequate assessment.

The censoring rules for PFS and DOR are given below in Table 1:

Table 1 Censoring Rules for PFS and DOR

| Situation | Date of Event<br>(Progression/Death due to<br>any cause) or Censored <sup>1</sup> | Event (Progression/Death due to any cause) Or Censored |
|---|---|---|
| Death due to any cause before<br>first assessment (or Death at<br>baseline or without any<br>adequate assessments) | Date of death | Event |
| No adequate baseline assessments and the participant has not died due to any cause (if the participant has died due to any cause follow the rules for death indicted at the top of the table) | Randomization date | Censored |
| No post-baseline assessments<br>and the participant has not<br>died due to any cause (if the<br>participant has died due to<br>any cause follow the rules for<br>death due to any cause<br>indicated at the top of the<br>table) | Randomization date | Censored |
| No adequate post-baseline assessment before start of new anticancer therapy | Randomization date | Censored |
| With post-baseline assessment<br>but no progression (or death<br>due to any cause) | Date of last 'adequate' assessment of response prior to any anti-cancer therapy | Censored |
| With adequate post-baseline assessment and new anticancer treatment started (prior to documented disease progression) <sup>2</sup> or death. | Date of last 'adequate'<br>assessment of response (on or<br>prior to starting anti-cancer<br>therapy) | Censored |
| Death due to any cause or progression after missing two | Date of last 'adequate' assessment of response <sup>3</sup> (prior to missed assessments): If the disease assessment is every 6 | Censored |

205801

| Situation | Date of Event<br>(Progression/Death due to<br>any cause) or Censored <sup>1</sup> | Event (Progression/Death due to any cause) Or Censored |
|---|---|---|
| or more scheduled assessments | weeks, a window of 91 days ([12=6*2] weeks + 7 day window) will be used to determine whether there is extended time without adequate assessment. If the time difference between PD/death due to any cause and last adequate disease assessment is more than 91 days, PFS will be censored at the last adequate disease assessment prior to PD/death due to any cause. For scans conducted after 49 weeks, a window of 175 days ([24=12*2]weeks + 7 day window) will be used to determine whether there is extended time without adequate assessment. | |
| Progression documented <sup>4</sup> | Date of assessment of progression | Event <sup>5</sup> |
| Death due to any casue <sup>4</sup> | Date of death | Event |

#### Notes:

For iPFS, iRECIST requires the confirmation of progression and uses the terms unconfirmed progressive disease (iUPD) and confirmed progressive disease (iCPD).

The progression event date (iPD date) to be used in the calculation of PFS per iRECIST should be the first date of documented iUPD provided that iCPD is confirmed at the next assessment.

<sup>&</sup>lt;sup>1</sup> Event or censored are based on confirmed responses.

<sup>&</sup>lt;sup>2</sup> If PD and New anti-cancer therapy occur on the same day assume the progression was documented first e.g., outcome is progression and the date is the date of the assessment of progression).

<sup>&</sup>lt;sup>3</sup> An adequate assessment is defined as an assessment where the response is (i)CR, (i)PR, (i)SD or any pseudo-progression (iUPD)

<sup>&</sup>lt;sup>4</sup> If both progression and Death due to any cause are documented then take the earliest date

<sup>&</sup>lt;sup>5</sup> If last response is iUPD and participant is still on treatment with no further response evaluation, then the participant will be censored at the last iUPD date for iPFS, else the participant will be considred for the event

205801

If more than one assessment is recorded as iUPD then the final occurrence prior to iCPD will be used. The exception to the rule would be when consecutive iUPDs followed by iCPD, the first occurrence of iUPDs in a row prior to iCPD will be used. For example, if a participant has iUPD at time points 1 and 2 and iCPD at time point 3, then iPD date would be the date of time point 1. If iUPD occurs, but is disregarded because of later iSD, iPR, or iCR, that iUPD date should not be used as the progression event date.

If progression is not confirmed and there is no subsequent iSD, iPR, or iCR, then the iUPD date will be used as iPD date in the following scenarios:

- Participant discontinues study intervention because the participant was judged not to be clinically stable
- Participant does not undergo further response assessments due to any reason (i.e., participant refusal, protocol non-compliance, or participant death)
- Next timepoint response of iUPD, and iCPD never occurs

# 7.2.2. Summary Measure

#### ORR

The number and percentage of participants with the BOR in the following response categories will be summarized: CR, PR,iCR,iPR. The corresponding exact 95% CI for ORR and iORR will also be provided. Participants with unknown or missing responses will be treated as non-responders, i.e., these participants will be included in the denominator when calculating percentages of response. A figure displaying maximum reduction in tumor size and listing of subject level responses will be generated.

#### DCR

The number and percentage of participants with the BOR in the following response categories will be summarized: CR, PR, SD, iCR,iPR, iSD. The corresponding exact 95% CI for DCR and iDCR will also be provided. Participants with unknown or missing responses will be treated as non-responders, i.e., these participants will be included in the denominator when calculating percentages of response.

#### **DOR**

The distribution of DOR will be summarized using the Kaplan-Meier method by treatment arm. The median, 25th and 75th percentiles of DOR will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method (Brookmeyer, 1982). Results from this will be descriptively summarised in tables and plotted, alogn with subject level listing of DOR.

#### **PFS**

The distribution of PFS for each treatment arm at will be estimated using the Kaplan-Meier method. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of PFS will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method (Brookmeyer, 1982). Results from this will be descriptively summarised in tables and plotted, along with subject level listing of PFS.

#### Milestone survival rate

The distribution of Milestone survival rate for each treatment arm at 12 months and 18 months will be estimated using the Kaplan-Meier method. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of OS will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method (Brookmeyer, 1982). Results from this will be descriptively summarised in tables and plotted, along with subject level listing of milestone survival.

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the ITT population, unless otherwise specified.

# 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. Key secondary endpoints, such as PFS, DOR and milstone survival rate will be analysed (see Section 7.2.4.1). Response rates estimates will be reported with 95% exact CI in the summary tables.

# 7.2.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

PFS, DoR

#### **Model Specification**

Hazard ratio for PFS and DoR and corresponding 95% confidence interval will be estimated
using the Cox's proportional hazard model stratified by the randomization factor(s) with
treatment arm as the sole explanatory variable.

#### **Model Checking & Diagnostics**

The proportional hazards assumption will be assessed using the following methods:

- Kaplan-Meier plot by treatment arm
- Plot of log(time) against log(-log(survival)) by treatment arm
- Plot of Schoenfeld residuals for treatment
- Evaluation of time-dependency of treatment effect by adding an interaction term of treatment and time in the Cox model. If the interaction term is significant (p< 0.05), it is considered that the proportional hazards assumption is violated.
- If one or more of the tests above demonstrates clear violation of the proportional hazards assumption, it is considered the proportional hazards assumption does not hold. Hazard ratio and corresponding 95% CI estimated from the Cox model will still be reported.
- Additional analysis of PFS and DoR are based on RMST, which does not require the proportional hazard assumption may be conducted.

Text below describes RMST Option 1: Commonly used pre-specified time-point:

Minimum of last event time in treat and control

Minimum of last observed time in treat and control

Time of clinical interest, e.g., 2 yrs.

SAS macro for calculation is available at: http://bcb.dfci.harvard.edu/~huno/computer-program/rmst2 ver003.sas

Text below describes RMST Option 2: The time interval should be between "larger than the maximum of smallest event time" and "smaller than the minimum of largest follow up time". R code for calculation is available at: http://onlinelibrary.wiley.com/doi/10.1111/biom.12384/abstract

### **Model Results Presentation**

Cox proportional hazard model results will be summarised in tables accounting for the stratification factors. The median, 25<sup>th</sup> and 75<sup>th</sup> percentiles of PFS/DoR will be estimated and corresponding 95% confidence intervals will be estimated using the Brookmeyer-Crowley method (Brookmeyer, 1982) and presented in tables. In addition Kaplan Mier figures will presented to show the distribution of PFS and DoR.

## Sensitivity and Supportive Analyses

If the proportional hazard assumption does not hold additional analysis based on RMST may be explored.

## **Endpoint / Variables**

ORR and DCR

### **Model Specification**

ORR and DCR will be compared between treatment arms using Cochran's Mantel Haenszel
test stratified by randomization factors. The exact 95% confidence interval for the difference
will be calculated.

## 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

# 8.1. Extent of Exposure

Extent of exposure to SOC and experimental arm will be summarized by Number of cycles, relative dose intensity and duration of exposure (see Section 12.6.2 for derivation details).

Relative dose intensity (RDI) is the percentage of the actual dose delivered relative to the intended dose. Relative dose intensity (RDI) is defined as (Actual cumulative dose delivered up to treatment discontinuation)/(Planned cumulative dose up to treatment discontinuation)\*100. The planned cumulative dose is the total dose that would be delivered, if there were no modification to dose or schedule. An RDI of 100% indicates that the drug was administered at the dose planned per protocol, without delay or reductions.

Treatment compliance is defined as (Actual cumulative dose/Scheduled cumulative dose)\*100. The scheduled dose accounts for any dose reductions, for example, if a participant had a dose reduction from 75 mg/m² to 60 mg/m², then the scheduled dose is 60 mg/m².

Summary statistics will be produced for extent of exposure.

Duration of Exposure in weeks is defined as (treatment stop date – treatment start date + 1) divided by 7.

For ITT Population, if subjects were randomized but did not receive any dose they will be counted as having zero duration of exposure. Duration of Study treatment will be plotted.

If the dose was not given at a particular visit, missed doses will be summarised and will include:

- number and percent of subjects with any missed doses. Each subject will only be counted once. The percentage will be based on "N".
- total number of missed doses (events).
- number and percent of subjects with any missed doses by category. Number of missed doses will be categorized as 0, 1, 2, 3 or more, and Not Evaluable. Not evaluable row is for subjects who did not receive any drug in any succeeding time period after the first dose. Each subject will only be counted once. The number from each row will add up to N. The percentage will be based on "N".
- number and percentage of missed doses (events) categorized by the reasons for missing a dose. Subject may be counted in multiple times in the same 'reason' row if the subject missed the dose multiple times for the same reason. Also, note that the same subject may be counted in multiple

reason rows, since they could have been missed a dose at different time points for different reasons. Therefore, the total number of events counted in different reasons must add up to the total number of missed doses (i.e. the number in the 2<sup>nd</sup> section of the table). The percentage will be based on the total number of missed doses (events).

Dose reductions will be summarised by treatment. The summary will include:

- number and percent of subjects with any reduction. Each subject will only be counted once. The percentage will be based on "N".
- total number of dose reductions (events).
- number and percent of subjects with any dose reduction by category. Number of dose reductions will be categorized as 0, 1, 2, 3 or more, and Not Evaluable. Not evaluable row is for subjects who did not receive any drug in any succeeding time period after the first dose. Each subject will only be counted once. The number from each row will add up to N. The percentage will be based on "N".
- number and percentage of dose reductions (events) categorized by the reasons. Subject may be counted in multiple times in the same 'reason' row if the subject had multiple dose reductions for the same reason. Also, note that the same subject may be counted in multiple reason rows, since their doses could have been reduced at different time points for different reasons. Therefore, the total number of events counted in different reasons must add up to the total number of dose reductions (i.e. the number in the 2<sup>nd</sup> section of the table). The percentage will be based on the total number of dose reductions (events).

Dose delays will be summarized by treatment and this will include:

- number and percent of subjects with any delay. Each subject will only be counted once. The percentage will be based on "N".
- total number of delays (events).
- number and percent of subjects with any dose delays by category. Number of dose delays will be categorized as 0, 1, 2, 3 or more, and Not Evaluable. Not evaluable row is for subjects who did not receive any drug in any succeeding time period after the first dose. Each subject will only be counted once. The number from each row will add up to N. The percentage will be based on "N".
- number and percent of dose delays (events) categorized by duration in days (e.g. 1-7, >=8 etc.). The percentages will be based on the total number of dose delays (i.e. the number from the 2<sup>nd</sup> section of the table). Subject may be counted in multiple times in the same 'duration' row if the subject had multiple dose delays for the same duration. Also, note that the same subject may be counted in multiple duration rows, since their doses could have been delayed at different time points for different lengths of time
- number and percentage of dose delays (events) categorized by the reasons. Subject may be counted in multiple times in the same 'reason' row if the subject had multiple dose delays for the same reason. Also, note that the same subject may be counted in multiple reason rows, since their doses could have been delayed at different time points for different reasons.

Therefore, the total number of events counted in different reasons must add up to the total number of dose delays (i.e. the number in the 2<sup>nd</sup> section of the table). The percentage will be based on the total number of dose delays (events).

Dose delay duration will be calculated as [start date of delayed dose - (start date of previous dose +21)]

If the infusions were stopped early and not completed it will be collected as incomplete infusions. Summary of Incomplete Infusion (by treatment) will include:

- number and percent of subjects with any incomplete infusion. Each subject will only be counted once. The percentage will be based on "N".
- total number of incomplete infusions (events).
- number and percent of subjects with any incomplete infusion by category. Number of incomplete infusion will be categorized as 0, 1, 2, 3 or more. Each subject will only be counted once. The number from each row will add up to N. The percentage will be based on "N".
- number and percentage of incomplete infusions (events) categorized by the reasons for stopping an infusion. Subject may be counted in multiple times in the same 'reason' row if the subject had incomplete infusion multiple times for the same reason. Also, note that the same subject may be counted in multiple reason rows, since they could have had incomplete infusions at different time points for different reasons. Therefore, the total number of events counted in different reasons must add up to the total number of incomplete infusions (i.e. the number in the 2<sup>nd</sup> section of the table). The percentage will be based on the total number of incomplete infusion (events).

If the infusions were intermittently interrupted but ultimately the infusion was completed it will be collected as infusion interruption. Summary of Infusion Interruptions (by treatment) will include:

- number and percent of subjects with any infusion interruptions. Each subject will only be counted once. The percentage will be based on "N".
- total number of infusion interruptions (events).
- number and percent of subjects with an infusion interruption by category. Number of infusion interruptions will be categorized as 0, 1, 2, 3 or more. Each subject will only be counted once. The number from each row will add up to N. The percentage will be based on "N".
- number and percentage of infusion interruptions (events) categorized by the reasons for interruption. Subject may be counted in multiple times in the same 'reason' row if the subject has infusion interruptions multiple times for the same reason. Also, note that the same subject may be counted in multiple reason rows, since they could have had infusion interruptions at different time points for different reasons. Therefore, the total number of events counted in different reasons must add up to the total number of infusion interruptions (i.e. the number in the 2<sup>nd</sup> section of

205801

the table). The percentage will be based on the total number of infusion interruptions (events).

All dose reductions, infusion interruptions and incomplete infusions, and dose delays will be listed separately by treatment.

# 8.2. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious adverse events (SAEs) and other significant AEs will be based on GSK Core Data Standards. Details on treatment emergent AEs are provided in Section 12.4.2. Dose modifications, dose interruptions, dose reduction dose delays will also be summarized and listed according to GSK Oncology Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

AEs will be coded using the standard MedDRA v.21.1. and grouped by system organ class. AEs will be graded by the investigator according to the NCI-CTCAE (version 5.0).

Summary of all Adverse Events and Drug related Adverse events by System Organ Class and Preferred Term and Maximum Grade will be reported. Summary of Grade 3-5 AEs and drug related Grade 3-5 AEs that occurred in ≥5% of participants will be provided by Overall frequency.

A summary of non-serious AEs that occurred in strictly 5% of the participants or above will be provided (no rounding for the percentage will be used in terms of 5% threshold, e.g. events with 4.9% incidence rate should not be included in this table).

A summary of number and percentage of participants with any adverse events by maximum grade will be produced. AEs will be sorted by PT in descending order of total incidence. The summary will use the following algorithms for counting the participant:

- **Preferred term row**: Participants experiencing the same AE preferred term several times with different grades will only be counted once with the maximum grade.
- **Any event row**: Each participant with at least one adverse event will be counted only once at the maximum grade no matter how many events they have.
- Summary of non-serious drug related adverse events by overall frequency by PT will be produced.

All AEs will be listed. Additionally, a listing of subject IDs for each individual AE will be produced. Listing of relationship of adverse event System Organ Class (SOC), Preferred term (PT) and verbatim text will be produced.

AEs with missing date of onset will be considered treatment-emergent.

# 8.3. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of

the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. The details of the planned displays are provided in Appendix 10: List of Data Displays.

AESI are currently defined as events of potential immunologic etiology (irAEs) (however this may change over time due to emerging data and analysies). Such events recently reported after treatment with other immune modulatory therapy include but not limited to:

| AE of | AE of Special | Preferred Term | System Organ | MedDRA |
|---|---|---|---|---|
| Special | Interest - Sub | (MedDRA | Class | Code |
| Interest | class | Version 21.1) | | |
| The followin | g is the synonyms o | f AEs of special interes | t will be combined u | inder the PT |
| | | special interest group | | ch other, |
| • | | or multiple AE of specia | · | 1 |
| Potential | Pneumonitis | Pneumonitis | Respiratory, | 10035742 |
| Immune- | | | thoracic and | |
| Mediated | | | mediastinal | |
| Disorders | | _ | disorders | |
| | | Dyspnoea | Respiratory, | 10013968 |
| | | | thoracic and | |
| | | | mediastinal<br>disorders | |
| | | Cough | | 10011224 |
| | | Cough | Respiratory,<br>thoracic and | 10011224 |
| | | | mediastinal | |
| | | | disorders | |
| | | Dyspnoea | Respiratory, | 10013971 |
| | | exertional | thoracic and | 10010371 |
| | | | mediastinal | |
| | | | disorders | |
| | | Rales | Respiratory, | 10037833 |
| | | | thoracic and | |
| | | | mediastinal | |
| | | | disorders | |
| | | Upper-airway | Respiratory, | 10070488 |
| | | cough syndrome | thoracic and | |
| | | | mediastinal | |
| | | | disorders | |
| | | Wheezing | Respiratory, | 10047924 |
| | | | thoracic and | |
| | | | mediastinal | |
| | | | disorders | |

| AE of<br>Special<br>Interest | AE of Special<br>Interest - Sub<br>class | Preferred Term<br>(MedDRA<br>Version 21.1) | System Organ<br>Class | MedDRA<br>Code |
|---|---|---|---|---|
| meerese | Class | Pneumonia | Infections and infestations | 10035664 |
| | | Pneumothorax | Respiratory,<br>thoracic and<br>mediastinal<br>disorders | 10035759 |
| | | Respiratory distress | Respiratory,<br>thoracic and<br>mediastinal<br>disorders | 10038687 |
| | | Hypoxia | Respiratory,<br>thoracic and<br>mediastinal<br>disorders | 10021143 |
| | Myocarditis | Myocarditis | | |
| | | Troponin Increased | | |
| | | Cardiac Ischemia | | |
| | | Myocardial<br>Infarction | | |
| | Colitis | Colitis | Gastrointestinal disorders | 10009887 |
| | | Diarrhea | Gastrointestinal disorders | 10012735 |
| | Hepatitis | Alanine<br>aminotransferase<br>increased | Investigations | 10001551 |
| | | Aspartate aminotransferase increased | Investigations | 10003481 |
| | | Blood alkaline<br>phosphatase<br>increased | Investigations | 10059570 |
| | | Blood bilirubin increased | Investigations | 10005364 |
| | | Hepatocellular injury | Hepatobiliary<br>disorders | 10019837 |
| | | Immnue-mediated hepatitis | Hepatobiliary<br>disorders | 10078962 |
| | | Hepatitis | Hepatobiliary<br>disorders | 10019717 |

| AE of | AE of Special | Preferred Term | System Organ | MedDRA |
|---|---|---|---|---|
| Special | Interest - Sub | (MedDRA | Class | Code |
| Interest | class | Version 21.1) | | |
| | | Hepatic function | Hepatobiliary | 10019670 |
| | | abnormal | disorders | |
| | | Transaminases increased | Investigations | 10054889 |
| | | Gamma-<br>glutamyltransferase<br>increased | Investigations | 10017693 |
| | Endocrinopathies | Hypophysitis | Endocrine<br>disorders | 10062767 |
| | | Hypopituitarism | Endocrine<br>disorders | 10021067 |
| | | Hypothyroidism | Endocrine<br>disorders | 10021114 |
| | | Hyperthyroidism | Endocrine<br>disorders | 10020850 |
| | | Hyperglycaemia | Metabolic and nutrition disorders | 10020635 |
| | Nephritis and<br>Renal Function | Renal impairment | Renal and urinary disorders | 10062237 |
| | | Acute kidney injury | Renal and urinary disorders | 10069339 |
| | | Blood creatinine increased | Investigations | 10005483 |
| | | Proteinurea | Renal and urinary disorders | 10037032 |
| | | Nephritis | Renal and urinary disorders | 10029117 |
| | | Pyelonephritis acute | Infections and infestations | 10037597 |
| | | Urinary retention | Renal and urinary disorders | 10046555 |
| | | Uninary incontinence | Renal and urinary disorders | 10046543 |
| | | Micturition urgency | Renal and urinary disorders | 10027566 |
| | Skin Adverse<br>Reactions | Rash | Skin and subcutaneous tissue disorders | 10037844 |

| AE of | AE of Special | Preferred Term | System Organ | MedDRA |
|---|---|---|---|---|
| Special | Interest - Sub | (MedDRA | Class | Code |
| Interest | class | Version 21.1) | | |
| | | Rash maculo- | Skin and | 10037868 |
| | | papular | subcutaneous | |
| | | | tissue disorders | |
| | | Rash Papular | Skin and | 10037876 |
| | | | subcutaneous | |
| | | | tissue disorders | |
| | | Pruritus | Skin and | 10037087 |
| | | | subcutaneous | |
| | | | tissue disorders | |
| | | Erythema | Skin and | 10015150 |
| | | | subcutaneous | |
| | | | tissue disorders | |
| | | Dermatitis | Skin and | 10012431 |
| | | | subcutaneous | |
| | | | tissue disorders | |
| | | Palmar-plantar | Skin and | 10033553 |
| | | erythrodysaesthesia | subcutaneous | |
| | | syndrome | tissue disorders | |
| | | Skin infection | Infections and | 10040872 |
| | | | infestations | |
| | | Skin ulcer | Skin and | 10040943 |
| | | | subcutaneous | |
| | | | tissue disorders | |
| | | Urticaria | Skin and | 10046735 |
| | | | subcutaneous | |
| | | | tissue disorders | |
| | | Vulvovaginal<br> | Reproductive | 10056530 |
| | | pruritus | system and | |
| | | Call livia | breast disorders | 40007000 |
| | | Cellulitis | Infections and | 10007882 |
| | | E - D - 21 - | infestations | 40052440 |
| | | Eye Pruritus | Eye disorders | 10052140 |
| | | Skin fissures | Skin and | 10040849 |
| | | | subcutaneous | |
| | Othor Irenevire | Danaraatitia | tissue disorders | 10022645 |
| | Other Immune- | Pancreatitis | Gastrointestinal | 10033645 |
| | Mediated | Lingso incressed | disorders | 10024574 |
| | Adverse Events | Lipase increased | Investigations | 10024574 |
| | | Amylase increased | Investigations | 10002016 |

205801

| AE of | AE of Special | Preferred Term | System Organ | MedDRA |
|---|---|---|---|---|
| Special | Interest - Sub | (MedDRA | Class | Code |
| Interest | class | Version 21.1) | | |
| | | Arthritis | Musculoskeletal and connective tissue disorders | 10003246 |
| Infusion-<br>Related<br>Reactions | Related | | General disorders and administration site conditions | 10008531 |
| | | Wheezing | Respiratory,<br>thoracic and<br>mediastinal<br>disorders | 10047924 |
| | | Pruritus | Skin and subcutaneous tissue disorders | 10037087 |
| | | Flushing | Vascular<br>disorders | 10016825 |
| | | Rash | Skin and subcutaneous tissue disorders | 10037844 |
| | | Hypotension | Vascular<br>disorders | 10021097 |
| | | Infusion related reaction | Injury, poisoning and procedural complications | 10051792 |
| | | Orthostatic hypotension | Vascular<br>disorders | 10031127 |

Summaries of the number and percentage of subjects with AESI will be provided for each type of event separately by preferred term and maximum grade.

Summary of Onset and Duration of the First Occurrence of AESI will also be produced.

#### 8.4. Deaths and Serious Adverse Events

All deaths will be summarised based on the number and percentage of participants. This summary will classify participants by time of death relative to the last dose of medication (>30 days or  $\leq$ 30 days) and primary cause of death (disease under study, SAE related to study treatment, or other). A supportive listing will be generated to provide participant-specific details on participants who died.

All SAEs will be tabulated based on the number and percentage of participants who experienced the event. The summary table will be displayed in descending order of total

205801

incidence by SOC and PT.Summary of Drug related SAE, fatal SAE, drug-related fatal SAE will also be produced

A study treatment-related SAE is defined as an SAE for which the investigator classifies the relationship to study treatment as "Yes". A worst-case scenario approach will be taken to handle missing data, i.e. the summary table will include events with the relationship to study treatment as 'Yes' or missing.

SAEs are included in the listing of all adverse events.

A listing of reasons for considering an SAE will be provided.

# 8.5. Adverse Events Leading to Discontinuation of Study Treatment and/or Withdrawal from the Study and Other Significant Adverse Events

The following categories of AEs will be summarized separately in descending order of total incidence by PT only and separate supportive listings will be generated with participant level details for those participants:

- AEs Leading to Discontinuation of Study Treatment
- AEs Leading to Withdrawal from the Study
- AEs Leading to Dose Interruptions
- AEs Leadings to Dose Reductions
- AEs Leading to Missed Doses

An AE leading to dose modification is an AE for which the action with respect to dosing is recorded as reduction or interruption of dose. AEs that lead to both a dose modification and a discontinuation of study treatment will only appear in the AEs leading to discontinuation of study treatment summary.

# 8.6. Pregnancies

While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE or SAE as described in the protocol. If subjects become pregnant while on the study, the information will be included in the narratives and no separate table or listing will be produced.

# 8.7. Clinical Laboratory Analyses

Laboratory grades will be reported using the Common Terminology Criteria for Adverse Events (CTCAE v5.0). The assessment of laboratory toxicities will examine the following laboratory tests performed by local laboratories:

| Laboratory Assessments | Parameters | | | |
|---|---|---|---|---|
| Hematology | RBC Indices | WBC count w | ith Differential | Platelets |
| | Hemoglobin | Neutrophils | | |
| | Hematocrit | Lymphocytes | | |
| | RBC count | Monocytes | | |
| | | Eosinophils | | |
| | | Basophils | | |
| Clinical Chemistry | BUNa | Potassium | Bilirubin | AST (SGOT) |
| | Creatinineb | Sodium | Total protein | ALT (SGPT) |
| | Glucose | Calcium | Albumin | Alkaline phosphatase |
| | LDH | | | |
| Coagulation | INR or PT | | | |
| _ | PTT/aPTT | | | |
| Cardiac Function | Troponin I or Troponin T | | | |
| Thyroid Function | Thyroid stimulating hormone | | | |
| , | Free T4 | J | | |
| | Free T3 (when | clinically indicate | d) | |
| Routine Urinalysis | Specific gravity | | | |
| | | | | (Note: routine urinalysis by |
| | method other than dipstick is acceptable, in accordance with local practice). | | | |
| Other Screening Tests | Hepatitis B surface antigen (HBsAg) | | | |
| | Hepatitis C (He | ep C antibody)º | | |
| | Serum β-hCG | Pregnancy test (fo | or women of child b | earing potential) |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase;  $\beta$ -hCG = beta-human chorionic gonadotropin; BUN = blood urea nitrogen; HBsAg = Hepatitis B surface antigen; RBC = red blood cells; SGOT = serum glutamic oxaloacetic transaminase; SGPT = serum glutamic pyruvic transaminase; T3 = triiodothyronine; T4 = thyroxine; WBC = white blood cells; INR = International Normalized Ratio; PT = Prothrombin Time; aPTT = Activated Partial Thromboplastin Time

- a. Required if local laboratory testing is available
- b. Creatinine clearance is also required to be calculated using the formula provided in Appendix 9 of the protocol.
- Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Hepatitis C RNA Test is optional with negative Hepatitis C antibody test.
- d. Coagulation factors (PT/INR and aPTT/PTT) should be tested as part of the screening procedures for all
  participants. Any participant receiving anticoagulant therapy should have coagulation factors monitored closely
  throughout the study

Change from baseline by scheduled visits will be summarised using mean, median, standard deviation, minimum, and maximum.

Summaries of worst case grade increase from baseline grade will be provided for all the lab tests that are gradable by CTCAE v5.0. These summaries will display the number and percentage of participants with a maximum post-baseline grade increasing from their baseline grade. Any increase in grade from baseline will be summarized along with any increase to a maximum grade of 3 and any increase to a maximum grade of 4. Missing baseline grade will be assumed as grade 0. In addition, the summary will include grade

205801

increase from baseline by scheduled visits. For laboratory tests that are graded for both low and high values, summaries will be done separately and labelled bi-direction, e.g. sodium will be summarized as hyponatremia and hypernatremia.

For lab tests that are not gradable by CTCAE v5.0, summaries of worst case changes from baseline with respect to normal range will be generated. Decreases to low, changes to normal or no changes from baseline, and increases to high will be summarized at each scheduled visit as well as for the worst case post-baseline. If a participant has a "Decrease to low" and an "Increase to high" during the same time interval, then the participant is counted in both the "Decrease to Low" category and the "Increase to High" category. In addition, the summary will include worst case changes from baseline with respect to normal range by scheduled visits.

Separate summary tables for hematology and chemistry laboratory tests will be produced.

Listing of Laboratory values of Potential Clinical Importance and listing of all laboratory values for any value of potential clinical importance will be produced

A separate listing of laboratory data with character values will also be provided. Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of participants with non-missing value at each visit.

Urinalysis Results will be summarised. Worst-case Urinalysis Results Post-Baseline Relative to Baseline will be summarised

A character lab value starting with '<X' or '>X' will be displayed in listings but will not be imputed with a numeric value thus will not be included for summaries.

# 8.8. Liver Function Analyses

Summaries of hepatobiliary laboratory abnormalities will be produced

Possible Hy's law cases are defined as any elevated (ALT  $\geq$ 3×ULN and overall bilirubin  $\geq$ 2×ULN (with direct bilirubin  $\geq$ 35% of total bilirubin, if direct bilirubin is measured) OR (ALT  $\geq$ 3×ULN and INR >1.5, if INR is measured). Note that INR measurement is not required and the threshold value stated will not apply to subjects receiving anticoagulants.

# 8.9. Other Safety Analyses

The analyses of non-laboratory safety test results including vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of subjects with non-missing value at each particular visit.

#### **Performance Status**

ECOG performance status will be summarized at baseline and each post-baseline scheduled visit. Summaries will use frequency and percentage of subjects at each planned assessment time.

A supporting listing will also be provided.

## Vital Signs

The following summaries will be provided for vital signs data:

- Summary of Changes in Heart Rate from Baseline
- Summary of Increases in Blood Pressure from Baseline
- Summary of Changes in Temperature from Baseline

The following listing will also be produced

• Listing of Vital Signs with Values of Potential Clinical Importance

The oncology standard categories for Heart Rate in bpm is:

• Heart Rate in bpm: 'Decrease to <60', 'Increase to >100'

The oncology standard categories for Systolic Blood Pressure in mmHg are:

- 'Any Grade Increase'
- 'Increase to Grade 2 (140-159)'
- 'Increase to Grade 3 (>=160)'

Note: 'Any Grade Increase' will be footnoted as Grade 0 (<120), Grade 1 (120-139), Grade 2 (140-159), Grade 3 (>=160).

The oncology standard categories for Diastolic Blood Pressure in mmHg are:

- 'Any Grade Increase'
- 'Increase to Grade 2 (90-99)'
- 'Increase to Grade 3 (>=100)'

Note: 'Any Grade Increase' will be footnoted as Grade 0 (<80), Grade 1 (80-89), Grade 2 (90-99), Grade 3 (>=100).

The oncology standard category 'Decrease to < 90' will be used for the Summary of decreases in Systolic Blood Pressure from Baseline.

The oncology standard categories of clinical concern for Temperature are:

• Temperature in C: 'Decrease to <=35', 'Increase to >= 38'

205801

#### **COVID-19 Assessments**

Confirmed, probable and suspected COVID 19 cases will be summarized and listed. Visits impacted by COVID-19 Pandemic will be summarized. Number of subjects with missed visits, site visits with one or more assessment missed, remote visit with no assessments missed and remote visit with one or more assessments missed will be summarized with primary reason for the impact.

## **Dose Limiting Toxicity**

For part 1 of the study, a listing of adverse events recorded as dose-limiting toxicities during the determinative period will be provided. Additionally, a summary of the number of patients experiencing DLTs will be provided.

## 9. PHARMACOKINETIC ANALYSES

# 9.1. Primary Pharmacokinetic Analyses

There are no primary pharmacokinetic analyses for this study.

# 9.2. Secondary Pharmacokinetic Analyses

## 9.2.1. Endpoint / Variables

### 9.2.1.1. **Drug Concentration Measures**

Details are included in Appendix 5: Data Display Standards & Handling Conventions (Section 12.5.3 Reporting Standards for Pharmacokinetic)

#### 9.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters for GSK3359609 and Docetaxel will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of Phoenix WinNonlin.

All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the GSK3359609 and Docetaxel concentration-time data, as data permits.

In addition to non-compartmental PK analysis, a preliminary population PK model developed from Phase I study 204691 may also be used to overlay observations from this study on PK model predictions (visual predictive check plots), and covariates may be explored to understand the variability in Cmax and Cmin parameters. To further support interpretation of PK data collected on 205801, PK information may be pooled with data from other trials and indications, including the phase I first-time-in-human (FTIH) study to develop and evaluate a basic structural PK model. This may be reported separately.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time 0 to the time of last quantifiable concentration will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed plasma concentration, determined directly from the concentration-time data. |
| Cmin | Minimum observed concentration |
| Ctau | Pre-dose (trough) drug concentration, where tau is the end of the dosing interval |

#### NOTES:

Additional parameters may be included as required.

## 9.2.2. Summary Measure

Plasma Concentration data will be summarised separately for GSK3359609 and Docetaxel. Corresponding listing of the plasma concentration values will also be produced. Individual plasma concentration-time plots by subject, mean concentration-

time plots and median concentration time plots will be produced for GSK3359609 and Docetaxel separately.

For each of these parameters for GSK3359609 and Docetaxel separately, the following summary statistics will be calculated for each treatment and presented separately: median, minimum, maximum, arithmetic mean, 95% confidence interval for the arithmetic mean, standard deviation, coefficient of variation (%CV = 100\*(sqrt (exp(SD²) - 1))) [NOTE: SD = SD of natural log (log<sub>e</sub>) transformed data]), geometric mean, 95% confidence interval for the geometric mean and standard deviation of natural logarithmically transformed data.

All PK parameters will be reported to at least 3 significant digits, but to no more significant digits than the precision of the original data.

All derived PK parameters will be listed.

## 9.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

# 9.2.4. Strategy for Intercurrent (Post-Randomization) Events

Not Applicable

### 10. SECONDARY ANALYSES

# 10.1. Immunogenicity Analyses

Serum samples will be collected and tested for the presence of antibodies that bind to GSK3359609 (ICOS agonist). These samples may also be tested for presence of antibodies that bind to Chinese Hamster Ovary (CHO) host cell proteins such as phospholipase B- like (PLBL2).

The actual date and time of each blood sample collection will be recorded. Details of blood sample collection (including volume to be collected), processing, storage, and shipping procedures are provided in the SRM.

Immunogenicity testing will occur in dosed subjects then analyzed, summarized descriptively and/or presented graphically.

Immunogenicity information will be listed by subject and a summary of the number of subjects that are negative and positive for the presence of the antibodies will be provided at each timepoint and overall for the subject. Drug tolerance of the assays will be taken into account in categorizing results at each timepoint as positive, negative, or inconclusive. A positive result at any timepoint means that the subject's overall category is positive.

# 10.2. Patient Reported Outcomes

Patient reported outcomes will be summarized in part 2 of the study.

# 10.2.1. Endpoint / Variables



# 10.2.2. Population of Interest

The PRO analyses will be based on the ITT population, unless otherwise specified.

# 10.2.3. Statistical Measures

# 10.2.3.1. Summary Measure







## 11. REFERENCES



Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, et al. Nivolumab versus docetaxel in advanced nonsquamous non–small-cell lung cancer. New England Journal of Medicine. 2015;373(17):1627-39.

Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, et al. Nivolumab versus docetaxel in advanced squamous-cell non-small-cell lung cancer. N Engl J Med. 2015; 373:123-35.

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics, 1982; 38:29-41.

Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumours: revised RECIST guidelines (version 1.1). Eur J Cancer. 2009; 45:228-47.



Gelman A, Carlin J, Stern H, et al. Bayesian Data Analysis. Third Edition. Boca Raton: CRC Press; 2013, page 41.

GlaxoSmiteKline Document Number 2017N337080\_02: A Phase II, Randomized, Openlabel Platform Trial Utilizing a Master Protocol to Study Novel Regimens Versus Standard of Care Treatment in NSCLC Participants.

Herbst RS, Baas P, Kim D-W, Felip E, Perez-Gracia JL, Han J-Y, et al. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small cell lung cancer (KEYNOTE-010): a randomised controlled trial. The Lancet. 2016;387(10027):1540-50.

Parmar M, Torri V, Stewart L. Extracting Summary Statistics to Perform Meta-Analysis of the Published Literature for Survival Endpoints. Statistics in Medicine. 1998; 17:2815-2834.

Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S et al. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. The Lancet Oncology. 2017 Mar 1;18(3):e143-e152. https://doi.org/10.1016/S1470-2045(17)30074-8

205801

Zhao L, Claggett B, Tian L, et al. On the restricted mean survival time curve in survival analysis. Biometrics. 2016; 72:215-221. Appendices

205801

# 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

There is no planned per protocol analysis for this study.

205801

# 12.2. Appendix 2: Schedule of Activities

# 12.2.1. Protocol Defined Schedule of Events

The Schedules of Activities can be found in the corresponding substudy appendix in Section 12.1

205801

# 12.3. Appendix 3: Assessment Windows

The visit assigned to the assessment as entered in the CRF (nominal visit) will be used for reporting.

# 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 12.4.1. Study Phases

Adverse events, serious adverse events, death and other safety domains will be assigned to the study phases defined below. Partial dates will be imputed into full dates, if applicable, for slotting data to the appropriate categories below. Flag variables (time in relation to study phase) indicating the study time periods will be added to the ADaM variable APHASE, and the treatment emergent AE flag will be created to ADAE variable TRTEMFL.

Assessments and events will be classified according to the time of occurrence relative to Study Treatment Start Date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 30 |
| | days |
| Post- | Date > Study Treatment Stop Date + 30 days |
| Treatment | |

For parameters where time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post- | Date > Study Treatment Stop Date |
| Treatment | |

#### 12.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to study treatment start date |
| Concomitant | Any medication that is not a prior |

#### **NOTES:**

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

205801

# 12.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | Non-serious AEs |
| Emergent | In general, all AEs with a start date after treatment are considered emergent regardless of AE start date is before or after treatment stop date. |
| | If AE onset date is on or after treatment start date & on or before treatment stop date + 30 days |
| | <ul> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date</li> <li>+ 30 days</li> </ul> |
| | <ul> <li>AE Start Date is missing</li> </ul> |
| | Serious AE/AESI |
| | <ul> <li>O If AE onset date is on or after treatment start date &amp; on or before treatment<br/>stop date + 30 days Study Treatment Start Date ≤ AE Start Date ≤ Study<br/>Treatment Stop Date + 30 days</li> </ul> |
| | <ul> <li>AE Start Date is missing</li> </ul> |
| | Missing AE Start Date will be imputed following rules in Section 12.7.2.1 for determining Treatment Emergent AEs. |

### NOTES:

- [If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.]
- If the study treatment stop date is missing, then the AE will be On-Treatment.
- Time of study treatment dosing and start[/stop] time of AEs should be considered, if collected.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

# 12.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently sup | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Compound | : Compound: GSK3359609, study: mid205801 |
| | Each IDMC interim and SAC relevant to eah substudy will be reported under mid205801 with a unique reporting effort. |
| <b>Analysis Datasets</b> | Analysis Datasets |
| <ul> <li>Analysis datasets will be created according to SDTM IG Version 3.2 &amp; ADaM IG Version 1.1.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for final SAC per substudy | |

## 12.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

205801

| Unscheduled Visits |
|---|
| All unscheduled visits will be included in listings. |
| Unscheduled visits will not be included in summary tables and/or figures, except for worst case summary tables and/or figures. |
| Descriptive Summary Statistics |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data N, n, frequency, % |
| Graphical Displays |
| Refer to IDSL Statistical Principals 7.01 to 7.13. |

# 12.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive<br>Summary Statistics,<br>Graphical Displays<br>and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Not Applicable. |
| NONMEM/PK/PD<br>File | Not applicable. |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to GUI_51487 |
| Descriptive<br>Summary Statistics,<br>Graphical Displays<br>and Listings | Graphical Displays Refer to GUI_51487 |

# 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time windowthe value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

## Study Day for Safety and PK

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - $\circ$  Ref Date < First Dose Date  $\rightarrow$  Study Day = Ref Date First Dose Date
  - Ref Date ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### Study Day for ITT

- Calculated as the number of days from Randomization Date:
  - Ref Date = Missing
  - o Ref Date < Randomization Date → Study Day = Ref Date Randomization Date
  - Ref Date ≥Randomization Date → Study Day = Ref Date Randomization Date + 1

→ Study Day = Missing

### **Change from Baseline**

- Change from Baseline = Post-Baseline Visit Value Baseline
- % Change from Baseline= 100 x (Post-Baseline Visit Value Baseline) / Baseline
- Maximum Increase/Decrease from Baseline = maximum (Increase/Decrease from Baseline)
- If either the Baseline or Post-Baseline Visit Value is missing, Change from Baseline and % Change from Baseline is set to missing

#### **Date of Response**

For post-baseline disease assessments, the date of response (PR or better) is assigned to the latest
date of disease assessments; for other response categories (SD [or Non-CR/Non-PD], NE, PD), the
date of response is assigned to the earliest date of disease assessments.

## **Date of New Anti-Cancer Therapy**

- Derived as the earliest date of new anti-cancer therapy, radiotherapy (where applicable) or surgical procedure (where applicable)
- Missing or partial dates will be imputed for derivation of new anti-cancer therapy following rules specified in Section 12.7.2.1.

#### **Duration and Elapsed Time**

- Durations (e.g., the duration of an adverse event, duration of exposure, etc.) are calculated as the stop date minus the start date plus one.
- For elapsed time (e.g., the time since initial diagnosis):
  - If the reference date is on or after the event date, then the elapsed time is the reference date minus the event date + 1
  - o If the reference date is before the event date, then the elapsed time is the reference date minus the event date
- For time to event (TTE) durations such as PFS

205801

- To report in months, divide the number of days by 30.4375
- To report in weeks, divide the number of days by 7
- To report in years, divide the number of days by 365.25.

These algorithms for time to event return decimal numbers and ignore the actual numbers of days in the months or years between start date and stop date. The "year" used in these algorithms is 365.25 days long, and the "month" is one twelfth of that year.

- For converting all other durations (e.g., duration of adverse events, duration of exposure, age) to weeks, months or years use the following:
  - To report the duration in weeks divide the number of days by 7
  - To report the duration in months use: (YEAR(stopdate + 1) YEAR(startdate)) \* 12 +
     (MONTH(stopdate + 1) month(startdate) 1) + (DAY(stopdate + 1) > = DAY(startdate))
  - To report the duration in years use:intck('year', startdate, stopdate + 1) (month(stopdate + 1) < month(startdate) or (month(stopdate + 1) = month(startdate) and day(stopdate + 1) < day(startdate)))

These algorithms return whole numbers for months and years, accurately accounting for the actual numbers of days in the months or years between the start date and the stop date.

# 12.6.2. Study Population

#### Demography

#### <u>Age</u>

- Age calculation will be based on Screening Date as the reference Date
- Birth date will be imputed as follows:

Any subject with a missing day will have this imputed as day '15'.

Any subject with a missing date and month will have this imputed as '30JUN'.

### **Extent of Exposure**

• The cumulative dose will be based on the formula:

Cumulative Dose = Sum of (the actual dose administered during each infusion)

• The relative dose intensity (%) is the infusion dose intensity divided by planned dose per week.

Relative Dose Intensity = (Cumulative Dose /Planned Dose)\*100

#### **Actual Treatment**

Participant's actual treatment will be derived from exposure data. If a participant's actual treatment is
the same as assigned treatment, actual treatment is the assigned treatment; if a participant received
treatment different from assigned treatment for the entire duration of treatment, actual treatment is
different from assigned treatment.

#### **Time since Initial Diagnosis**

- Calculated as the number of [Days] from the Date of Initial Diagnosis:
  - First Dose Date = Missing → Elapse Time = Missing
  - Date of Initial Diagnosis = Completely/partially Missing → Elapse Time = Missing
  - Otherwise → Elapse Time = First Dose Date Date of Initial Diagnosis + 1

205801

## 12.6.3. Safety

| Adverse Events | | |
|---|---|---|
| AE'S OF Special Interest | | |
| Refer to Section 8.2 | | |
| Duration of AE | | |
| Calculated as the number of [days] from AE Start Date to AE Stop Date: | | |
| | AE Start Date = Missing | → Elapse Time = Missing |
| | AE Stop Date = Missing | → Elapse Time = Missing |
| | Otherwise | → Elapsed Time = AE Stop Date – AE Start Date + 1 |

## **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
- Example 3: 0 Significant Digits = '< x' becomes x − 1</li>

# 12.6.4. Patient Reported Outcomes (PRO)



205801 CCI














205801

## 12.7. Appendix 7: Reporting Standards for Missing Data

### 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>A participant will be considered to have completed the study if the participant dies during the study treatment period or follow-up period, whichever is sooner, or is still in followup at the time of the final analysis.</li> <li>A participant will be considered to have withdrawn from the study if the participant has not died and is lost to follow-up, has withdrawn consent, at the investigator's discretion is no longer being followed or if the study is closed/terminated.</li> <li>Participants who discontinue will not be replaced in this study. All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays. However where necessary, display macros may impute dates as temporary variables for sorting data in listings only. In addition, partial dates may be imputed for 'slotting' data to study phases (see Section 12.4.1) or for specific analysis purposes as outlined below.</li> </ul> |
| | <ul> <li>Imputed partial dates will not be used to derive study day, time to onset or<br/>duration (e.g., time to onset or duration of adverse events), or elapsed time<br/>variables (e.g., time since diagnosis). In addition, imputed dates are not used for<br/>deriving the last contact date in overall survival analysis dataset.</li> </ul> |
| Adverse Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following conventions:</li> </ul> |
| | <ul> <li>Missing start day</li> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> </ul> </li> </ul> |

| Element | Reporting Detail | |
|---|---|---|
| | | <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing stop day | Last day of the month will be used. |
| | Missing stop day and month | No Imputation |
| | Completely missing start/end date | No imputation |
| Concomitant Medications/ Blood Supportive | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: | |
| Products | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year) |
| | Missing end day and month | A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date | No imputation |

| Element | Reporting Detail |
|---|---|
| New Anti-Cancer<br>Therapy/<br>Radiotherapy/<br>Surgical<br>Procedures for<br>Efficacy<br>Evaluation (e.g.,<br>response rate,<br>time to event) | <ul> <li>Completely missing start dates will remain missing, with no imputation applied;</li> <li>Partial start dates will be imputed using the following convention: <ul> <li>If both month and day are missing, no imputation will be applied;</li> <li>If only day is missing: <ul> <li>If the month of partial date is the same as the month of last dosing date, minimum of (last dosing date + 1, last day of the month) will be used for the day;</li> <li>If the month of partial date is the same as the month of last disease assessment and the last disease assessment is PD, minimum of (last date of disease assessment + 1, last day of the month) will be used for the day;</li></ul></li></ul></li></ul> |
| ECG | <ul> <li>Missing baseline values are assumed to have baseline value &lt;450 for<br/>QTc</li> </ul> |

205801

### 12.8. Appendix 8: Values of Potential Clinical Importance

To identify values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v [5.0]) will be used to assign grades for laboratory parameters including clinical chemistry, hematology, liver function tests, QTc (Fridericia's) values, LVEF and vital signs (heart rate, blood pressure, temperature).

Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings.

205801

# 12.9. Appendix 9: Abbreviations & Trade Marks

## 12.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| ADA | Anti-drug antibodies |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CR | Complete Response |
| DOB | Date of Birth |
| DOR | Duration of Response |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FA | Final Analysis |
| FDA | Food and Drug Administration |
| FDAAA | · · |
| GSK | Food and Drug Administration Clinical Results Disclosure Requirements GlaxoSmithKline |
| (i)CR | |
| (i)PR | Complete Response as per (i)RECIST 1.1 |
| iUPD | Partial Response as per (i)RECIST 1.1 |
| iCPD | Unconfirmed Progressive Disease as per iRECIST 1.1 |
| (i)SD | Confirmed Progressive Disease as per iRECIST 1.1 |
| (i)PFS | Stable Disease as per (i)RECIST 1.1 |
| (i)ORR | Progression free survival as per (i)RECIST 1.1 |
| (i)DOR | Overall response rate as per (i)RECIST 1.1 Duration of Response as per (i)RECIST 1.1 |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | |
| IDSL | Independent Data Monitoring Committee Integrated Data Standards Library |
| IMMS | Integrated Data Standards Library International Modules Management System |
| ITT | International Modules Management System Intent-To-Treat |
| IV | Intravenous |
| IWRS | Interactive web response system |
| LFT | Liver function test |
| LVEF | Left ventricular ejection fraction |
| NCI-CTCAE | National Cancer Institute - Common Terminology Criteria for Adverse Events |
| NSCLC | Non-small-cell lung cancer |
| CCI | Tron on any our or |
| ORR | Overall Response Rate |
| OS | Overall Survival |
| PA | Primary Analysis |
| PCI | Potential Clinical Importance |
| . 51 | r otential official importance |

205801

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| PD | Progressive Disease |
| PFS | Progression Free Survival |
| PDMP | Protocol Deviation Management Plan |
| CCI | |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PR | Partial Response |
| PRO | Patient-reported outcome |
| CCI | |
| CCI | |
| QoL | Quality of Life |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RECIST | Response evaluation criteria in solid tumours |
| SAC | Statistical Analysis Complete |
| SD | Stable Disease |
| SDTM | Study Data Tabulation Model |
| SoC | Standard of Care |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

## 12.9.2. Trademarks

| Trade | marks of the GlaxoSmithKline<br>Group of Companies |
|-------|----------------------------------------------------|
| NONE | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonLin |

205801

### 12.10. Appendix 10: List of Data Displays

### 12.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|--------------------------|-------------|------------|
| Study Population | 1.1 to 1.23 | |
| Efficacy | 2.1 to 2.12 | 2.1 to 2.6 |
| Safety | 3.1 to 3.34 | 3.1 to 3.2 |
| Pharmacokinetic | 4.1 to 4.4 | 4.1 to 4.6 |
| Patient Reported Outcome | 5.1 to 5.12 | 5.1 to 5.6 |
| Section | List | ings |
| ICH Listings | 1 to | 35 |
| Other Listings | 36 t | o 44 |

### 12.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Section 12.11: Example Mock Shells for Data Displays.

| Section | Figure | Table |
|--------------------------|--------|---------|
| Safety | | SAFE_Tn |
| Patient Reported Outcome | PRO_Fn | PRO_Tn |

#### 12.10.3. Deliverables

| Delivery | Description |
|----------|----------------------------------------------------|
| Part 1 | Futility analysis |
| IDMC | Independent Data Monitoring Committee Open session |
| PA | Primary Analysis |
| FA | Final Statistical Analysis Complete |

205801

# 12.10.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | ITT/Safety | ES8 | Summary of Subject Status and Reason for Study Withdrawal | ICH E3, FDAAA, EudraCT Part 1 is based on Safety population Part 2 is based on ITT population | PART1,<br>IDMC/PA.<br>FA,(Headline) |
| 1.2. | Safety | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | PART1, IDMC/<br>PA. FA,<br>(Headline) |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | PART1, IDMC/<br>PA. FA, |
| 1.4. | ITT/Safety | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| 1.5. | Screened | SP1 | Summary of Study Populations | IDSL | PART1, PA. FA, |
| Protoc | ol Deviation | | | | |
| 1.6. | ITT/Safety | DV1 | Summary of Protocol Deviations | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population Separate the page by important and non-important deviations | PART1, PA. FA, |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphics | | | | |
| 1.7. | ITT/Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT Include baseline stratification factors Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA,<br>(Headline) |
| 1.8. | ITT/Safety | DM11 | Summary of Age Ranges | EudraCT Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| 1.9. | ITT/Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| Prior a | nd Concomitan | t Medications | | | |
| 1.10. | ITT/Safety | MH1 | Summary of Past Medical Conditions | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| 1.11. | ITT/Safety | MH1 | Summary of Current Medical Conditions | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| 1.12. | ITT/Safety | CM1 | Summary of Concomitant Medications | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | PART1, PA. FA, |
| Diseas | e Characteristic | cs | | <u> </u> | |
| 1.13. | ITT | DC1 | Summary of Disease Characteristics at Initial Diagnosis | ICH E3 | IDMC/ PA. FA, |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.14. | ITT | DC2 | Summary of Disease Characteristics at Baseline | ICH E3 Add definitions for progression and recurrence | IDMC/ PA. FA,<br>(Headline) |
| 1.15. | ITT | MD1 | Summary of Metastatic Disease at Screening | | IDMC/ PA. FA, |
| 1.16. | ІТТ | LA1 | Summary of Disease Burden at Baseline | ICH E3 | IDMC/ PA. FA, |
| Anti-Ca | ncer Therapy | | | | |
| 1.17. | ITT/Safety | AC1 | Summary of Prior Anti-Cancer Therapy | IDSL Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| 1.18. | ITT/Safety | CM1 | Summary of Prior Dictionary Coded Anti-Cancer Therapy | IDSL Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| 1.19. | ITT/Safety | AC3 | Summary of Number of Prior Anti-Cancer Therapy Regimens | IDSL Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| 1.20. | ITT/Safety | FAC1 | Summary of Follow-up Anti-Cancer Therapy | IDSL Part 1 is based on Safety population Part 2 is based on ITT population | PART1, PA. FA |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Surgica | I/Medical Proc | edures | | | |
| 1.21. | ITT/Safety | OSP1 | Summary of Prior Surgical Procedures | IDSL Part 1 is based on Safety population Part 2 is based on ITT population | PART1, IDMC/<br>PA. FA, |
| Substar | nce Use | | | | |
| 1.22. | ITT | SU1 | Summary of Substance Use | IDSL | IDMC/ PA. FA, |
| Follow- | Follow-up | | | | |
| 1.23. | ITT | FAC2 | Summary of Duration of Follow-up | | PA. FA, |

205801

# 12.10.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Respor | ises | | | | |
| 2.1. | ITT /Safety | RE1a | Summary of Confirmed Investigator-Assessed Best Response (RECIST1.1) | Add rows for DCR (CR+PR+SD), Odds ratio for DCR, 95% CI and p-Value Part 1 is based on Safety population Part 2 is based on ITT population | PART1, PA.<br>FA,(Headline) |
| 2.2. | ITT | RE1a | Summary of Confirmed Investigator-Assessed Best Response (iRECIST Criteria) | Add rows for DCR<br>(CR+PR+SD), Odds ratio for<br>DCR, 95% CI and p-Value | PA. FA, |
| 2.3. | ІТТ | RE2 | Summary of Investigator Assessed Response Rate with confirmation (RECIST1.1 Criteria) by Stratification Factors | <ul> <li>Histology (squamous vs. non squamous) and line of PD(L)1 therapy (1st vs. 2nd line).</li> <li>Add Count and percentages for DCR ( CR+PR+SD)</li> </ul> | PA. FA, |
| 2.4. | ITT | RE2 | Summary of Investigator Assessed Response Rate with confirmation (iRECIST Criteria) by Stratification Factors | Add Count and percentages for DCR (CR+PR+SD) | PA. FA, |

| Time-to | -event Endpoi | nts | | | |
|---|---|---|---|---|---|
| 2.5. | ITT | TTE3 | Summary of Kaplan-Meier Estimates of Progression-Free<br>Survival | Using RECIST1.1 followed by iRECIST on next page Do not report p-values | PA.<br>FA,(Headline) |
| 2.6. | ITT | TTE3 | Summary of Kaplan-Meier Estimates of Overall Survival | Do not report p-values | PA.<br>FA,(Headline) |
| 2.7. | ITT | TTE6 | Summary of Kaplan-Meier Estimates of Overall Survival at 12 and 18 Months | | PA. FA, |
| 2.8. | ITT | TTE1 | Summary of Kaplan-Meier Estimates of Duration of Response in Subjects with Objective Response | Page by RECIST1.1 then iRECIST | PA.<br>FA,(Headline) |
| 2.9. | ITT | TTE4 | Summary of Cox Proportional Hazards Regression Model for<br>Overall Survival | Remove p-value column Include a row for predictive probability of Phase 3 success as the last segment | PA.<br>FA,(Headline) |
| 2.10. | | | Model Diagnostic SAS outputs from Cox Proportional Hazards model for Overall Survival | RTF format of SAS results output | PA. FA, |
| 2.11. | ITT | TTE4 | Summary of Cox Proportional Hazards Regression Model for Overall Survival (Sensitivity Analysis for Adjusting the Impact of COVID 19) | | PA. FA, |
| 2.12. | ITT | TTE4 | Summary of Cox Proportional Hazards Regression Model for<br>Progression Free Survival | Remove p-value column Page by RECIST 1.1 then iRECIST | PA. FA, |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Respor | Responses | | | | |
| 2.1. | ITT /Safety | RE1a | Summary of Confirmed Investigator-Assessed Best Response (RECIST1.1) | Add rows for DCR (CR+PR+SD), Odds ratio for DCR, 95% CI and p-Value Part 1 is based on Safety population Part 2 is based on ITT population | PART1, PA.<br>FA,(Headline) |
| 2.2. | ITT | RE1a | Summary of Confirmed Investigator-Assessed Best Response (iRECIST Criteria) | Add rows for DCR<br>(CR+PR+SD), Odds ratio for<br>DCR, 95% CI and p-Value | PA. FA, |
| 2.3. | ITT | RE2 | Summary of Investigator Assessed Response Rate with confirmation (RECIST1.1 Criteria) by Stratification Factors | <ul> <li>Histology (squamous vs. non squamous) and line of PD(L)1 therapy (1st vs. 2nd line).</li> <li>Add Count and percentages for DCR ( CR+PR+SD)</li> </ul> | PA. FA, |
| 2.4. | ITT | RE2 | Summary of Investigator Assessed Response Rate with confirmation (iRECIST Criteria) by Stratification Factors | Add Count and percentages for DCR (CR+PR+SD) | PA. FA, |

| Time-to | -event Endpoi | nts | | | |
|---|---|---|---|---|---|
| 2.5. | ITT | TTE3 | Summary of Kaplan-Meier Estimates of Progression-Free Survival | Using RECIST1.1 followed by iRECIST on next page Do not report p-values | PA.<br>FA,(Headline) |
| 2.6. | ITT | TTE3 | Summary of Kaplan-Meier Estimates of Overall Survival | Do not report p-values | PA.<br>FA,(Headline) |
| 2.7. | ITT | TTE6 | Summary of Kaplan-Meier Estimates of Overall Survival at 12 and 18 Months | | PA. FA, |
| 2.8. | ITT | TTE1 | Summary of Kaplan-Meier Estimates of Duration of Response in Subjects with Objective Response | Page by RECIST1.1 then iRECIST | PA.<br>FA,(Headline) |
| 2.9. | ITT | TTE4 | Summary of Cox Proportional Hazards Regression Model for<br>Overall Survival | Remove p-value column Include a row for predictive probability of Phase 3 success as the last segment | PA.<br>FA,(Headline) |
| 2.10. | | | Model Diagnostic SAS outputs from Cox Proportional Hazards model for Overall Survival | RTF format of SAS results output | PA. FA, |
| 2.11. | ITT | TTE4 | Summary of Cox Proportional Hazards Regression Model for<br>Overall Survival (Sensitivity Analysis for Adjusting the Impact of<br>COVID 19) | | PA. FA, |
| 2.12. | ITT | TTE4 | Summary of Cox Proportional Hazards Regression Model for<br>Progression Free Survival | Remove p-value column Page by RECIST 1.1 then iRECIST | PA. FA, |

205801

# 12.10.6. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Respon | ise | | | | |
| 2. | ITT | RE8a | Investigator-Assessed Maximum Percent Reduction from Baseline in Tumor Measurement (RECIST1.1) | | PART1, PA.<br>FA, |
| Time-to | -Event Endpoi | nts | | | |
| 2.2. | ITT | TTE10 | Graph of Kaplan Meier Survival Curves for Progression Free Survival with 95% Confidence Band | Page by RECIST1.1 then iRECIST. | PA.<br>FA,(Headline) |
| 2.3. | ITT | TTE10 | Graph of Kaplan Meier Curves for Overall Survival | Include line at 12 months and 18 months to approximate the rate and 95% CI. | PA.<br>FA,(Headline) |
| 2.4. | ITT | TTE10 | Graph of Kaplan Meier Curves for Duration of Response in Subjects with Objective Response | Page by RECIST1.1 then iRECIST | PA. FA, |
| 2.5. | ITT | TTE11 | Forest Plot of r Overall Survival by Subgroup | | PA.<br>FA,(Headline) |
| 2.6. | ITT | TTE11 | Forest Plot of Progression Free Survival by RECIST1.1. by Subgroup | | PA. FA, |

205801

# 12.10.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE5B | Summary of Treatment Emergent Adverse Events by System<br>Organ Class and Preferred Term and Maximum Grade | | PART1, PA. FA, |
| 3.2. | Safety | OAE07 | Summary of Treatment Emergent Adverse Events by Preferred Term and Maximum Grade | | PART1, PA. FA,<br>(Headline) |
| 3.3. | Safety | AE13 | Treatment Emergent Adverse Events Overview | Include Any AE, AEs related to study treatment, leading to permanent discontinuation of study treatment, leading to dose reduction, leading to dose interruption/delay, Any SAE, SAEs related to study treatment, Fatal SAEs, Fatal SAEs related to study treatment Add an additional row to indicate frequency and percentage of Treatment Related AE's of grade 3+4+5 | PART1, PA. FA,<br>(Headline) |
| 3.4. | Safety | AE3 | Summary of Common (>=5%) Grade 3-5 Treatment Emergent Adverse Events by Overall Frequency | | PART1, PA. FA,<br>(Headline) |
| 3.5. | Safety | OAE01 | Summary All Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term and Maximum Grade | | PART1, PA. FA, |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | Safety | AE15 | Summary of Common (>=5%) Non-serious Treatment Emergent<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Participant and Occurrences) | | PART1, PA. FA, |
| 3.7. | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 3-5 Treatment Emergent Adverse Events by Overall Frequency | | PART1, PA. FA, |
| 3.8. | Safety | AE3 | Summary of Non-Serious Drug-Related Treatment Emergent Adverse Events by Overall Frequency | | PART1, PA. FA, |
| Advers | e Events of Sp | ecial Interest | | | · |
| 3.9. | Safety | OAE01 | Summary of Adverse Event or Condition of Special interest by Preferred Term and Maximum Grade | | PART1, PA. FA, |
| 3.10. | Safety | ESI2a | Summary of Onset and Duration of the First Occurrence of AE of Special Interest | | PART1, PA. FA, |
| Serious | and Other Sig | nificant Adverse l | Events | | · |
| 3.11. | Safety | AE16 | Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | PART1, PA. FA,<br>(Headline) |
| 3.12. | Safety | AE3 | Summary of Treatment Emergent Adverse Events Leading to Permanent Discontinuation of Study Treatment by Preferred Term | | PART1, PA. FA, |
| Deaths | | | | | |
| 3.13. | Safety | DTH1a | Summary of Deaths | IDSL | PART1, PA. FA,<br>(Headline) |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Chemistry | <i>y</i> | | | |
| 3.14. | Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | PART1, PA. FA, |
| 3.15. | Safety | OLB9C | Summary of Worst Case Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 | PART1, PA. FA, |
| 3.16. | Safety | OLB11C | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | PART1, PA. FA, |
| Labora | t <mark>ory: Hematolo</mark> | gy | | | |
| 3.17. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | PART1, PA. FA, |
| 3.18. | Safety | OLB9C | Summary of Worst Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 | PART1, PA. FA, |
| 3.19. | Safety | OLB11C | Summary of Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | PART1, PA. FA, |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Urinalysis | <b>.</b> | | | |
| 3.20. | Safety | LB1 | Summary of Urinalysis Results | ICH E3 | PART1, PA. FA, |
| 3.21. | Safety | OUR1B | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | PART1, PA. FA, |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.22. | Safety | OLIVER1 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | PART1, PA. FA, |
| Vital Si | gns | l | | | 1 |
| 3.23. | Safety | OVT1B | Summary of Changes in Vital Signs from Baseline | | PART1, PA. FA, |
| Exposu | re/Dose Modifi | ications | | | |
| 3.24. | Safety | SAFE_T1 | Summary of Exposure to Treatment | Add a footnote defining the "Cycle" | PART1, PA. FA,<br>(Headline) |
| 3.25. | Safety | ODMOD4 | Summary of Missed Doses by Component | Exclude the last segment "Number of Subjects with Missed Doses by Planned Time" | PART1, PA. FA, |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.26. | Safety | ODMOD1 | Summary of Dose Reductions | Exclude the last segment "Number of Subjects with Dose Reduction by Planned Time". Count number of participants and total number of reductions if either component is reduced. Summarise details on number and reason by component in separate rows | PART1, PA. FA, |
| 3.27. | Safety | ODMOD3 | Summary of Dose Delays | Exclude the last segment "Number of Subjects with Dose Delays by Planned Time". Count number of participants and total number of delays if either component is delayed. Summarise details on number, duration and reason by component in separate rows | PART1, PA. FA, |
| 3.28. | Safety | ODMOD9 | Summary of Incomplete Infusions | Exclude the last segment "Number of Subjects with Incomplete Infusions by Planned Time" | PART1, PA. FA, |
| 3.29. | Safety | ODMOD16 | Summary of Infusion Interruptions | Exclude the last segment" Number of Subjects with Infusion Interruptions by Planned Time" | PART1, PA. FA, |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Perform | nance Status | | | | |
| 3.30. | Safety | PS1A | Summary of ECOG Performance Status | ICH E3 | PART1, PA. FA, |
| lmmun | ogenecity | | | | • |
| 3.31. | Safety | IMM1 | Summary of Positive Immunogenecity Results | | PART1, PA. FA, |
| COVID- | 19 Assessmen | ts | | | |
| 3.32. | Safety | PAN1 | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events | | PART1, PA. FA, |
| 3.33. | Safety | PAN3 | Summary of COVID-19 Symptoms for Subjects with COVID-19 Adverse Events | | PART1, PA. FA, |
| Dose L | imiting Toxicity | / (DLT | | | |
| 3.34. | DLT<br>Evaluable | AE19 | Summary of Dose-Limiting Toxicities during the Determinative Period (DE Phase) | | PART1 |

205801

# 12.10.8. Safety Figures

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposure | | | | | |
| 3.1. | Safety | OEX12 | Plot of Duration of Study Treatment | | PA. FA, |
| Laborat | ory | | | | |
| 3.2. | Safety | Liver9 | Scatter Plot of Maximum Bilirubin versus Maximum ALT – eDISH | | PA. FA, |

205801

## 12.10.9. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | | | | | |
| 4.1. | PK | PK01 | Summary of GSK3359609 Plasma Concentration Time Data | IDSL | FA, SAC |
| 4.2. | PK | PK01 | Summary of Docetaxel Plasma Concentration Time Data | IDSL | FA, SAC |
| 4.3. | PK | PK06 | Summary of Derived GSK3359609 Pharmacokinetic Parameters (non-transformed and log-transformed) | IDSL | FA, SAC |
| 4.4. | PK | PK06 | Summary of Derived Docetaxel Parameters (non-transformed and log-transformed) | IDSL | FA, SAC |

205801

# 12.10.10. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | | | | | · |
| 4.1. | PK | PK16a | Individual GSK3359609 Plasma Concentration-Time Plot by Subject (Linear and Semi-Log) | IDSL | FA, SAC |
| 4.2. | PK | PK16a | Individual Docetaxel Plasma Concentration-Time Plot by Subject (Linear and Semi-Log) | IDSL | FA, SAC |
| 4.3. | PK | PK17 | Mean GSK3359609 Concentration-Time Plots (Linear and Semi-log) | IDSL | FA, SAC |
| 4.4. | PK | PK17 | Mean Docetaxel Concentration-Time Plots (Linear and Semilog) | IDSL | FA, SAC |
| 4.5. | PK | PK18 | Median GSK3359609 Concentration-Time Plots (Linear and Semi-log) | IDSL | FA, SAC |
| 4.6. | PK | PK18 | Median Docetaxel Concentration-Time Plots (Linear and Semilog) | IDSL | FA, SAC |

205801

# 12.10.11. Patient Reported Outcomes Tables

| Patient | Patient Reported Outcome: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

| Patient | Patient Reported Outcome: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

| Patient | Patient Reported Outcome: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | - | | | - <b>/-</b> |

205801

## 12.10.12. Patient Reported Outcomes Figures



205801

# 12.10.13. ICH Listings

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subje | ect Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | Part1, IDMC/<br>PA. FA, |
| 2. | ITT/Safety | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | Part1, IDMC/<br>PA. FA, |
| 3. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | Part1,IDMC/ PA.<br>FA, |
| 4. | ITT | TA1 | Listing of Planned and Actual Treatments | IDSL | PA. FA, |
| Proto | col Deviations | | | | - |
| 5. | ITT/Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | Part1, PA. FA, |
| 6. | ITT/Safety | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | Part1, IDMC/<br>PA. FA, |
| Demo | graphic and Bas | seline Characteristic | s | | |
| 7. | ITT/Safety | DM2 | Listing of Demographic Characteristics | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | Part1, IDMC/<br>PA. FA, |

| ICH: I | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 8. | ITT/Safety | DM9 | Listing of Race | ICH E3 Part 1 is based on Safety population Part 2 is based on ITT population | Part1, IDMC/<br>PA. FA, |
| Prior | and Concomitan | t Medications | | | |
| 9. | ITT/Safety | CP_CM3 | Listing of Prior/Concomitant Medications | IDSL Part 1 is based on Safety population Part 2 is based on ITT population | Part1, PA. FA, |
| 10. | ITT/Safety | MH2 | Listing of Past/Current Medical Conditions | Oncology specific template to be used Part 1 is based on Safety population Part 2 is based on ITT population | Part1, IDMC/<br>PA. FA, |
| Expo | sure and Treatm | ent Compliance | | | |
| 11. | Safety | OEX8a | Listing of Exposure to Docetaxel | ICH E3 | PA. FA, |
| 12. | Safety | OEX8b | Listing of Exposure to GSK3359609 | ICH E3 | Part1, PA. FA, |
| 13. | Safety | COMP2 | Listing of Overall Compliance | | Part1, IDMC/<br>PA. FA, |
| Dose | Modifications | | | | |
| 14. | Safety | ODMOD10A | Listing of Dose Reductions | Exclude Cycle | Part1, PA. FA, |

| ICH: L | _istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 15. | Safety | ODMOD17A | Listing of Infusion Interruptions | Exclude Cycle | Part1, PA. FA, |
| 16. | Safety | ODMOD14A | Listing of Incomplete Infusions | Exclude Cycle Day | Part1, PA. FA, |
| 17. | Safety | ODMOD12A | Listing of Dose Delays | Exclude Cycle Day | Part1, PA. FA, |
| 18. | Safety | ODMOD13A | Listing of Missed Doses | Exclude Cycle | Part1, PA. FA, |
| Resp | onse | | | | |
| 19. | ITT/Safety | LA5 | Listing of Investigator Assessed Lesion Assessments (RECIST 1.1 Criteria) | Include Target Lesions,Non-Target Lesions and New Part 1 is based on Safety population Part 2 is based on ITT population | Part1, PA. FA, |
| 20. | ITT | LA5 | Listing of Investigator Assessed Lesion Assessments (iRECIST Criteria) | Include Target Lesions,Non-Target Lesions and New Lesions | PA. FA, |
| 21. | ITT/Safety | RE5 | Listing of Investigator Assessed Responses with confirmation (RECIST 1.1 Criteria) | Part 1 is based on Safety population Part 2 is based on ITT population | Part1, PA. FA, |
| 22. | Safety/ITT | RE5 | Listing of Investigator Assessed Responses with confirmation (iRECIST Criteria) | Part 1 is based on Safety population Part 2 is based on ITT population | Part1, PA. FA, |
| Adve | rse Events | | | | |
| 23. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | Part1, PA. FA, |
| 24. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | Part1, PA. FA, |
| 25. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | Part1, PA. FA, |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse Events of Special Interest | | | | | |
| 26. | Safety | AE8 | Listing of AE of Special Interest | | Part1, PA. FA, |
| Serious and Other Significant Adverse Events | | | | | |
| 27. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse<br>Event | ICH E3 | Part1, PA. FA, |
| 28. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | Part1, PA. FA, |
| Deaths | | | | | |
| 29. | Safety | DTH3 | Listing of Deaths | ICH E3 | Part1, PA. FA, |
| Hepatobiliary (Liver) | | | | | |
| 30. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | Part1, PA. FA, |
| 31. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | Part1, PA. FA, |
| All Laboratory | | | | | |
| 32. | Safety | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | Part1, PA. FA, |
| 33. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | Part1, PA. FA, |
205801

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Performance Status | | | | | |
| 34. | Safety | PS5A | Listing of Performance Status | | Part1, PA. FA, |
| Dose-Limiting Toxicities | | | | | |
| 35. | DLT Evaluable | MTD_DLDL1 | Listing of Dose-Limiting Toxicities (DLT) during the determinative period (DE Phase) | | Part1 |

205801

## 12.10.14. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Diseas | e Characteristi | cs | | | |
| 36. | ITT | DC3 | Listing of Disease Characteristics at Initial Diagnosis | | IDMC/ PA. FA, |
| 37. | ITT | DC4 | Listing of Disease Characteristics at Screening | | IDMC/ PA. FA, |
| Anti-Ca | ancer Therapy | I | | | |
| 38. | ITT | AC6 | Listing of Prior Anti-Cancer Therapy | | IDMC/ PA. FA, |
| 39. | ITT | AC7 | Listing of Prior Anti-Cancer Radiotherapy | | IDMC/ PA. FA, |
| 40. | ITT | FAC3 | Listing of Follow-Up Anti-Cancer Therapy | | PA. FA, |
| Surgica | al Procedures | 1 | | 1 | |
| 41. | ITT | OSP3 | Listing of Prior Surgical Procedures | | PA. FA, |
| lmmun | ogenecity | | | | |
| 42. | Safety | IMM2 | Listing of Immunogenicity Results | | PA. FA, |
| PK | • | 1 | | | 1 |
| 43. | PK | PK07 | Listing of Pharmacokinetic Concentration-Time Data by Analyte | IDSL | PA. FA, |
| 44. | PK | PK13 | Listing of Derived Pharmacokinetic Parameters by Analyte | IDSL | PA. FA, |

205801

## 12.11. Appendix 11: Example Mock Shells for Data Displays

Data Display Specification will be made available on request.

205801

# 12.12. Appendix 12: SDAC REPORTING PLAN

GSK Protocol 205801 - GSK3359609 ENTREE Study

Version: Final

Date: 20 February 2020

#### 13. INTRODUCTION

This document, the SDAC Reporting Plan for GSK Protocol 205801, describes SDAC's proposal for the initial content and structure of Independent Data Monitoring Committee (IDMC) reports. It includes general statistical analysis conventions and a detailed proposed table of contents. Mock tables, figures, and listings are provided in a companion document, the SDAC Sample Report.

This document is the final version of SDAC Reporting Plan for GSK Protocol 205801. The drafted version (and the companion *SDAC Sample Report*) has been distributed to the DMC and GSK prior to the first IDMC meeting for review and discussion.

The IDMC, SDAC, and GSK recognize that for the IDMC to effectively execute their responsibility to oversee the safety of subjects enrolled in the study, they will require interim reporting that meets their needs as those needs evolve over the duration of the studies. As such, this proposal is intended as a general guide for the content and structure of initial reports to be produced by SDAC for the IDMC and it is not intended to either limit the scope of the analyses the IDMC may request or to require a particular form or structure for an analysis. It is understood that the IDMC will have the final authority to specify, on an ongoing basis, the content and structure of the reports they receive.

#### 13.1. References to External Documents

Where this document excerpts or references external documents, the following versions have been used:

- *IDMC Charter* (Version 001, dated December 19, 2018)
- SDAC Sample Report (dated September 20, 2016)
- Study Protocol (205801 Amendment #1 dated September 20, 2018)
- *Study RAP* (Statistical Analysis Plan Reporting and Analysis Plan dated December 13, 2018)
- AESI Listing (GSK3359609 AESI list FINAL 03Apr19 Version 1.xlsx)

# 13.2. OVERVIEW OF ANALYSES SPECIFIED IN THE IDMC CHARTER

SDAC will prepare both open session and closed session reports containing summaries of safety and/or efficacy data for data review meetings starting when adequate data are available. Data review meetings will be held at least every 6 months, but more frequent meetings may be held.

As described in the *IDMC Charter*, the IDMC will review the following data for study 205801: "Summarized unblinded safety data including AEs, SAEs, immune-related adverse events (irAEs), adverse events of special interest (AESI), and laboratory data for all active substudies. Summarized unblinded efficacy data primary endpoints and selected

205801

secondary endpoints such as ORR, PFS, etc. Note that if a substudy or treatment arm has been discontinued, this data will not require further review."

As such, the safety reports from each of the studies will contain, at a minimum, analyses of all adverse events, serious adverse events (including deaths and SUSARs if recorded), withdrawals due to adverse events, laboratory values, and available efficacy data. All IDMC recommendations will be made based on a review of the totality of evidence.

As stated in the *IDMC Charter*, Section 3.5, "At the planned interim analyses in the 205801 study, the IDMC may make the recommendation to halt an individual substudy or study treatment arm (other than SoC) due to safety concerns and/or lack of efficacy." Additionally, the IDMC may recommend the discontinuation of an experimental regimen based on the totality of evidence to protect the safety, in relation to efficacy, of participating subjects. As such, closed session reports will include primary interim efficacy measures. Open session reports will omit these analyses to preserve blinding.

The details of these reports are described in Section 13.4.

#### 13.3. GENERAL SDAC REPORTING CONVENTIONS

#### 13.3.1. Sample Report

The separate document titled *SDAC Sample Report* provides an example of IDMC report content and format for a single, fictitious protocol based on simulated data. This fictitious protocol is patterned after a typical cardiovascular study, and therefore the example analyses are not tailored to the specifics of this study's design.

Actual reports for the GSK 205801 study will include initial content as proposed in detail in Section 4 below.

In the remainder of this document, references in doubled square brackets are to pages of the *Sample Report* (e.g., [[Figure ACCR-1, p. 18]]).

#### 13.3.2. Open and Closed Session Reports

SDAC will produce Closed Session and Open Session versions of IDMC reports.

Closed Session reports will include analyses of all relevant data by treatment group. These reports will be only for review by the IDMC and will not be shared with other parties prior to database lock for the study. Treatment groups will be identified by single-letter codes with assignment of codes to treatment arms provided to the IDMC members in a separate document. Codes will be consistent between reports over the life of the trial.

Open session reports will include displays of aggregate data only (no treatment group information) and so will be fully blinded. Open session reports will also *exclude* efficacy

analyses and any additional analyses requested by the IDMC on the basis of their unblinded review. Open session reports will be provided to all open session participants, including the IDMC and GSK.

#### 13.3.3. General Analysis Conventions

Reports will include analyses of all randomized subjects restricted to (1) post-randomization event data and (2) baseline and post-randomization data from other sources. In particular, analyses will exclude subjects that are screened but not randomized and will exclude any adverse events occurring prior to randomization.

All analyses will be performed on an intention-to-treat basis with subjects analyzed as randomized irrespective of adherence to treatment. In particular, analyses will include data collected for subjects who discontinue treatment but remain on study.

In general, for follow-up data collected on a per-visit basis (*e.g.*, laboratory measurements and vital signs) that include a visit code and a visit date, analyses by scheduled visit will use the visit code rather than applying a windowing algorithm to the visit date, and unscheduled visits will be excluded. Analyses that aggregate postbaseline data (*e.g.*, plots showing numbers of subjects who *ever* had a post-baseline, abnormal value for a laboratory measurement) will use all post-baseline measurements, whether scheduled or unscheduled.

#### 13.3.4. Graphical Conventions

The primary mode of presentation in SDAC IDMC reports is graphical; most presented graphics have supporting back-up tables in the Supporting Material section of the report (see SDAC Sample Report, p. 74).

Categorical data will be presented as simple or stacked bar charts where the height of the bar or bar segment, respectively, represents the percent of subjects in a particular category (e.g., see Gender, Race, and NYHA Class in [[Figure DEMO-1, p. 28]]). Continuous data will be presented as boxplots where the bottom whisker, bottom edge of the box, horizontal line through the box, top edge of the box, and top whisker indicate the 5th, 25th (Q1), 50th (median), 75th (Q3), and 95th percentiles of the data, respectively, and a plotting symbol indicates the mean (e.g., see Age and Left Ventricular Ejection Fraction in [[Figure DEMO-1, p.28]]).

Time-to-event data will be presented as Kaplan-Meier plots of cumulative incidence (e.g., [[Figure ENDPT-3, p. 71, top panel]]). In the Closed Session Reports, treatment comparisons for time-to-event analyses across different endpoints or for a single endpoint across different subgroups will be presented as forest plots showing point estimates and 95% confidence intervals (CIs) for hazard ratios (HRs), as in [[Figure ENDPT-4, p. 73]].

A section of Supporting Material [[p. 74]] will contain back-up tables for the graphical displays of the previous chapters. These tables will be cross-referenced to and from the corresponding graphical pages.

#### 13.3.5. P-values

In the closed session report, p-values for treatment comparisons will be provided for most post-baseline analyses. These p-values should be viewed as screening tools, rather than formal hypothesis tests, as no adjustment will be made for multiple tests performed. Given the large number of tests to be considered, it would be expected that a number of p-values will appear statistically significant (<0.05) simply by chance.

Except where otherwise noted, p-value calculations for continuous or ordered categorical data will use the nonparametric Wilcoxon-rank sum test (or Kruskal-Wallis test as appropriate), p-values for dichotomous and unordered categorical data will use Pearson's chi-square test without continuity correction, and p-values for time-to-event data will use a log-rank test.

#### 13.3.6. Use of Listings when Data Are Limited

The study is expected to enroll 105 patients in the initial treatment arms, but early IDMC reports may include displays incorporating limited data on a small number of randomized patients. The detailed table of contents below and the Sample Report companion to this document assume a sufficient amount of data to support the use of graphical and tabular summaries. However, for initial reports where data for some displays are very limited, listings may be more appropriate and useful. SDAC will exercise its judgment in its use of graphics and tables versus listings in initial reports. On an ongoing basis, the IDMC, in consultation with SDAC, will evaluate the relative suitability of listings alone, summaries supplemented by listings, and summaries alone to communicate the results of interim analyses, and SDAC will adapt its reporting accordingly.

#### 13.3.7. Considerations for Analysis of Interim Data

IDMC reports will be based on data from interim snapshots of the study database and other interim sources of data. These sources are likely to include so-called "dirty" data: records that are incomplete, inconsistent, entered in error, not yet adjudicated or coded, and otherwise under query. As a general approach, SDAC will include all available data in interim analyses, implementing reasonable conventions to resolve inconsistencies and handle incomplete records while utilizing statistical approaches that are robust in the face of errors.

Detailed conventions for handling dirty data will be documented in the introductory material of IDMC reports, but general approaches will include:

- Removing implausible or impossible values or assuming an appropriate unit conversion (e.g., height of 180 inches)
- Using simple hierarchical definitions for potentially contradictory sources of information (e.g., calculating a death date using the adjudicated result if available and falling back on dates included in the clinical endpoint dataset, from fatal adverse event records in the adverse event dataset, etc.)
- Presenting uncoded adverse events (AEs) in a separate category using the investigator-supplied verbatim term in tables and listings

- Completing partial dates using a sensible algorithm (e.g., middle of month if day is missing; middle of year if day and month are missing; with appropriate truncation for dates known or likely to be postrandomization)
- Use of statistical techniques that are robust in the face of gross errors such as use of quantile-based descriptive statistics (medians, quartiles, and 5<sup>th</sup> and 95<sup>th</sup> percentiles) and non-parametric tests (Wilcoxon)

#### 13.4. PROPOSED DETAILED TABLE OF CONTENTS

The list below represents the proposed content for the Closed Session Report. The Open Session Report will have similar content (with analyses for randomized trials performed in aggregate only without respect to treatment group) but will exclude certain analyses as indicated above.

In the following, references are given to representative examples of content in the *Sample Report*, though analyses in actual reports may be presented in a different form (*e.g.*, listings in place of summaries where data are limited). Example graphics are presented with two treatment groups, though graphics for GSK 205801 may be modified to include three or more contrasts as applicable (see *Sample Report*, *Chapter A3*, p. 127).

#### 13.4.1. Accrual and Study Status

[See the Sample Report Chapter 1 for illustrative examples.]

- Subject accrual over time by treatment arm (line plot, with bar graph by month) [[Figure ACCR-1, p. 18]]
- Site accrual over time (line plot, with bar graph by month) [[Figure ACCR-2, p. 19]]
- Geographic distribution of randomized subjects and randomizing sites (bar graph, table) [[Figures ACCR3-4, pp. 20-21]]
- Accrual by stratification factors (squamous vs non-squamous, 1<sup>st</sup> vs 2<sup>nd</sup> line of PD(L) 1 therapy) (bar graph)
- Subject treatment status, and reasons for IP discontinuation (bar graphs) [[Figure STAT-1, p. 23]]
- Subject study/completion status, and reasons for early study termination (bar graphs) [[Figure STAT-1, p.
   23]]
- Protocol violation/deviations (listing)

#### 13.4.2. Baseline Characteristics

[See the Sample Report Chapter 2 for illustrative examples.]

- Demographics [age, gender, race, ethnicity] (boxplot, bar graphs) [[Figure DEMO-1, p. 28]]
- Medical history (bar graph) [[Figure MDHX-1, p. 29]]
- Concomitant medication use at baseline by coded category (table)

- Vital signs [temperature, pulse rate, respiratory rate, blood pressure] (boxplots) [[Figure VITB-1, p. 30]]
- Physical measurements [height, weight, BMI] (boxplots) [[Figure VITB-1, p. 30]]
- Baseline labs [[Figure LABB-1, p. 31]]

#### 13.4.3. Adverse Events

[See the Sample Report Chapter 3 for illustrative examples.] Serious adverse events:

- Listing of deaths
- Overview [any SAE, any SAE possibly related to study treatment, SAE leading to IP and/or study discontinuation, any fatal SAE] (bar graph) [[Figure SAE-1, p. 33]]
- Tabulation by SOC and High Level Term/Preferred Term (tables) [[Table SAETAB, p. 35]]
- Listing of SAEs by subject (listing showing treatment group, subject ID, sex, age, country, randomization date, start and end day of event relative to randomization and treatment periods, MedDRA preferred

term, action taken with respect to study drug) [[Figure AELISTING-1, p. 38]]

Adverse events (whether serious or non-serious) leading to study drug discontinuation:

- Overview (AEs leading to treatment discontinuation, study withdrawal, dose interruptions/reductions) (bar graph) [[Figure AE-1, p. 39]]
- AE frequency by MedDRA SOC (stacked bars indicating max severity) [[Figure AE-2, p. 40]]
- Most common AEs [by MedDRA PT/HLT] (stacked bars indicating max severity) [[Figure AE-3, p. 41]]
- AEs with a nominally significant treatment difference (closed session only) [[Figure AE-4, p. 42]]
- Tabulation of by SOC and PT/HLT (tables) [[Table AETAB, p. 43] Immune-related adverse events (irAEs)
  - irAEs as described in Section 7.2.1.1 and Table 8 (p. 41) of the *Study Protocol* (bar graphs) [[similar to Figure AE-2, p.40]]

Adverse events of Special Interest (bar graphs) [[similar to Figure AE-2, p. 40]]

- Subclasses of AEs provided to SDAC by GSK in AESI LISTING: 

   Pneumonitis, colitis, hepatitis, endocrinopathies, nephritis and renal function, skin adverse reactions, other immune-mediated adverse events (see AESI LISTING for full specifications)
- Infusion-related reactions o (see AESI LISTING for full specifications)

#### 13.4.4. Central Laboratory Measures

Open session reports will omit all laboratory results that may unblind the study sponsor; SDAC will communicate with GSK to establish any lab parameters to be omitted.

[See the Sample Report Chapter 4 for illustrative examples.] General laboratory presentation:

- Summary page for each set of tests showing the percent above and/or below thresholds, as appropriate, for each test in the set (bar charts, with stacked bars for categorical assessments and for LFT elevations categorized by multiples of ULN) [[Figure LFTABN-1, p.49]]
- Each laboratory measure by scheduled visit [[Figure LFT-1, p. 50]]: o For most lab tests, multiple panels: measurements at each visit (boxplot), change from baseline (boxplot), percent of subjects above and/or below thresholds (ULN, LLN, or other clinically defined values of concern) at each visit (bar graph)
  - For ordered categorical results (*e.g.*, some urinalysis assessments):
    stacked bars indicating the percent of subjects in each category at each visit
     Categories of laboratory measures displayed using above presentation:
    - Hematology
    - Clinical chemistry
    - Urinalysis

#### 13.4.5. Other Follow-up Measures

[See the Sample Report Chapter 5 for illustrative examples.]

- Vital signs [body temperature, pulse rate, respiratory rate, systolic and diastolic blood pressure] (box plots by visit, with change from baseline) [[Figure VIT-1, p. 60]]
- Physical measurements [weight, BMI] (boxplots) [[Figure VIT-3, p. 62]]
- Physical exam [clinically significant changes since previous visit] (listing)
- ECG interpretation (bar graph by visit) [[Figure ECG-1, p. 63]]
- ECG data [QT, QTcF RR, GR, PR, QRS] (box plots by visit, with change from baseline) [[Figure ECG-2, p. 64]]

#### 13.4.6. Efficacy and Interim Analyses

As specified in Section 3.1 of the *Study RAP*, formal interim analyses will be conducted by SDAC and presented to the IDMC in closed session. These analyses will be triggered after approximately 45 total observed events in the combined experimental and SoC arms, with a minimum of 18 events in the experimental arm.

[See the Sample Report Chapter 6, Study Endpoints, pp. 69-72 for illustrative examples] Primary Efficacy Parameters:

• Predictive probability of Phase III study success for each treatment arm as described in Section 10.5.1 of the *Study Protocol* — if triggered by events.

205801

#### Key secondary Efficacy Parameters

- All-cause mortality (overall survival) (Cumulative mortality, forest plot) [[ENDPT-3, p. 71; ENDPT-4, p.72]]
- Kaplan-Meier estimates of milestone survival rates at 12 and 18 months (forest plot) [[similar to ENDPT4, p. 72]]

Note: Shells can be found here:

https://biostat.wiscweb.wisc.edu/wp-content/uploads/sites/1008/2019/05/Sample\_Report\_Closed\_20160920.pdf

### Signature Page for 205801 TMF- 1714066 v 3.0

| Reason for signing: Approved | Name: PPD Role: A Date of signature: 06-Mar-2021 20:43:40 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD<br>Role: A<br>Date of signature: 08-Mar-2021 16:38:04 GMT+0000 |

Signature Page for TMF-1714066 v3.0